CLINICAL TRIAL: NCT04436120
Title: TREATMENT RESISTANCE FOLLOWING ANTI-CANCER THERAPIES (TRANSLATE)
Brief Title: Treatment Resistance Following Anti-cancer Therapies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lack of enrollment that has been compounded by the global COVID-19 pandemic. There were no safety and/or efficacy concerns involved in the decision to stop enrollment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A9001502; TRANSLATE (Other: Alias Study Number); 2018-003612-45 (EudraCT Number)
Record Dates: First submitted 2020-06-09; First posted 2020-06-17 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Disease Progression
Keywords: Non Small Cell Lung Cancer; Renal Cell Carcinoma; HR+ HER2- Breast Cancer; Castrate-Resistant Prostate Cancer; Germline mutated BRCA, HER2- Breast Cancer
MeSH Terms: conditions — Disease Progression; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor biopsy and blood draw (Other): Tumor biopsy and blood draw
  Interventions: Procedure: De novo tumor tissue biopsy; Procedure: Research blood draws

INTERVENTIONS:
Procedure: De novo tumor tissue biopsy — De novo tissue biopsy performed following disease progression
Procedure: Research blood draws — Blood biospecimens collected following disease progression

SUMMARY:
The TRANSLATE study aims to better understand why tumors become resistant to standard anti-cancer therapies.

New tumor biopsy and blood samples are collected after disease progression on standard-of-care anti-cancer treatment and compared to the initial (archival) tumor biopsy sample taken from the same patient.

Annotated reports of results from clinical Next Generation Sequencing (NGS) gene panel tests of both tumor and blood are sent directly from the testing lab to the study physician for discussion with the patient during the study.

Patients may participate in interventional treatment clinical trials at the same time as participating in the TRANSLATE study.

Primary data will be publicly available after the study to support further research.

DETAILED DESCRIPTION:
Background: Development of new cancer treatments requires better understanding of why tumors develop resistance to standard-of-care (SOC) therapies. However, post-progression tumor biopsies are not routinely collected, limiting the tissue available to characterize mechanisms of treatment resistance. The TRANSLATE clinical study is specifically designed to address these critical gaps.

Trial design: TRANSLATE is a global, multicenter, translational study designed to collect and compare archival pre-treatment tumor tissue with paired de novo tumor and blood samples obtained following disease progression on SOC therapies, targeting therapeutically important areas of cancer biology.

Eligible Tumor Type and Most Recent SOC Therapy:

* Non-small-cell lung and Anti-PD-1/-L1 monotherapy
* Non-small-cell lung and Anti-PD-1/-L1 + platinum
* Clear cell renal cell carcinoma and Anti-PD-1/-L1 monotherapy
* Clear cell renal cell carcinoma and Doublet anti-PD-1/-L1 + anti-CTLA-4
* Clear cell renal cell carcinoma and Pembrolizumab + axitinib
* Clear cell renal cell carcinoma and Avelumab + axitinib
* HR+ HER2- breast and Palbociclib + hormonal therapy
* germline mutated BRCA breast and Olaparib or talazoparib monotherapy
* Castration-resistant prostate and Enzalutamide
* Castration-resistant prostate and Abiraterone + prednisone

Eligibility criteria include adults with locally advanced or metastatic tumors; radiographic evidence of progressive disease during the most recent SOC regimen; sufficient archival tumor tissue; and a post-progression tumor lesion that is safely accessible for a new biopsy.

The results from clinical NGS panel testing may help inform subsequent treatment plan or identification of relevant interventional clinical trials.

Patients are enrolled after disease progression on SOC and before change in treatment and participate in 3 study visits within approximately 3 months.

Next-generation sequencing results from analysis of tumor tissue and blood will be returned to the study physician and patient for review at a subsequent study visit within this timeframe.

The primary endpoint is the change in frequency of gene alterations between pre-treatment and post-progression tumor biopsies. Secondary endpoints address prioritized scientific hypotheses specific to each target area of biology and indication.

Primary data will be publicly available after the study to support further research.

Sponsored by Pfizer Inc.; EudraCT: 2018-003612-45.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of locally advanced (primary or recurrent) or metastatic solid tumors treated as follows:
* Non small cell lung carcinoma (NSCLC) monotherapy: Disease progression (PD) on 1st line monotherapy anti PD-1/ L1.
* NSCLC combination: PD on 1st line anti PD-1/ L1 plus standard doublet platinum containing regimen; or PD on 1st-line anti-PD-1/-L1 plus standard doublet platinum-containing regimen followed by continuation of single agent anti-PD-1/-L1).
* Renal cell carcinoma (RCC) with clear cell component: PD on 2nd line monotherapy anti PD-1/ L1; or PD on 1st line combination of doublet anti-PD-1/ L1 with anti-CTLA-4; or PD on 1st-line combination of avelumab with axitinib or pembrolizumab with axitinib.
* HR+ HER2 adenocarcinoma of the breast: PD on 1st line combination of doublet palbociclib with hormonal therapy.
* Castrate resistant adenocarcinoma of the prostate: PD on enzalutamide monotherapy.
* Castrate resistant adenocarcinoma of the prostate: PD on abiraterone in combination with prednisone.
* germline mutated BRCA (gBRCAm), HER2- breast cancer: PD on a PARP inhibitor monotherapy in patients previously treated with chemotherapy in the neoadjuvant, adjuvant, or metastatic setting.
* Radiographic evidence of PD, including the target lesion being subjected to biopsy for the study, on the most recent regimen that requires a change in anti-cancer treatment.

Exclusion Criteria:

* Tumor biopsy taken from a bone or an irradiated target lesion.
* Discontinuation of current or most recent anti cancer therapy due to toxicity and not progressive disease.
* Initiation of new anti-cancer therapy after disease progression prior to planned biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (16):
  - Southern Cancer Center, P.C., Daphne, Alabama
  - Southern Cancer Center, PC, Mobile, Alabama
  - Alaska Urological Institute dba Alaska Clinical Research Center, Anchorage, Alaska
  - Arizona Oncology Associates, PC-HOPE, Tucson, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - The Oncology Institute of Hope Innovation, Glendale, California
  - The Oncology Institute of Hope Innovation, Long Beach, California
  - UCI Medical Center-Chao Family Comprehensive Cancer Center, Orange, California
  - The Oncology Institute of Hope Innovation, Santa Ana, California
  - Sansum Clinic, Santa Barbara, California
  - Sansum Clinic, Solvang, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - ICRI-Administrative and Supplies Only, Whittier, California
  - Woodlands Medical Specialists PA, Pensacola, Florida
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Argentina (4):
  - Clínica Viedma S.A., Viedma, Río Negro Province
  - Sanatorio de la Mujer, Rosario, Santa Fe Province
  - Hospital Britanico de Buenos Aires, CABA
  - Centro de Educacion Medica e Investigaciones Clinicas"Norberto Quirno" CEMIC, Ciudad Autónoma de Bs As
- Belgium (5):
  - Grand Hôpital de Charleroi - Site Notre Dame, Charleroi
  - AZ Maria Middelares, Ghent
  - UZ Gent, Ghent
  - Hôpital de Jolimont, Haine-Saint-Paul
  - Clinique Saint-Pierre Ottignies, Ottignies
- France (6):
  - Centre Jean Perrin, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Centre Hospitalier Louis Pasteur, Colmar
  - CHU Henri Mondor, Créteil
  - Hôpital La Croix du Sud, Quint-Fonsegrives
  - Institut Jean Godinot, Reims
  - Hopital Bégin, Saint-Mandé
- Royal Cornwall Hospital, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A9001502

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 38 participants were enrolled into 7 cohorts. The Safety Analysis (SA) population included 36 participants who had de novo biopsy or research blood draw performed.
Groups:
- Cohort 1: Non-small Cell Lung Carcinoma (NSCLC) Monotherapy: Progressive disease on 1st line monotherapy anti-programmed cell death receptor 1 or programmed cell death ligand 1 (anti-PD-1/-L1).
- Cohort 2: NSCLC Combination: Progressive disease on 1st line anti-PD-1/-L1 plus standard doublet platinum-containing regimen; or progressive disease on 1st line anti-PD-1/-L1 plus standard doublet platinum-containing regimen followed by continuation of single agent anti-PD-1/-L1.
- Cohort 3: Renal Cell Carcinoma (RCC) With Clear Cell Component: Progressive disease on 2nd line monotherapy anti-PD-1/-L1; or progressive disease on 1st line combination of doublet anti-PD-1/-L1 with anti-CTLA-4; or progressive disease on 1st line combination of avelumab with axitinib or pembrolizumab with axitinib.
- Cohort 4: Hormone Receptor+Human Epidermal Growth Factor Receptor 2 - Adenocarcinoma of the Breast: Progressive disease on 1st line combination of doublet palbociclib with hormonal therapy.
- Cohort 5: Castrate-resistant Adenocarcinoma of the Prostate: Progressive disease on enzalutamide monotherapy.
- Cohort 6: Castrate-resistant Adenocarcinoma of the Prostate: Progressive disease on abiraterone in combination with prednisone.
- Cohort 7: Germline Mutated BRCA (gBRCAm) HER2- Adenocarcinoma of the Breast: Progressive disease on a poly ADP-ribose polymerase (PARP) inhibitor monotherapy in participants previously treated with chemotherapy in the neoadjuvant, adjuvant, or metastatic setting.
Period: Overall Study
Arm/Group | Cohort 1: Non-small Cell Lung Carcinoma (NSCLC) Monotherapy | Cohort 2: NSCLC Combination | Cohort 3: Renal Cell Carcinoma (RCC) With Clear Cell Component | Cohort 4: Hormone Receptor+Human Epidermal Growth Factor Receptor 2 - Adenocarcinoma of the Breast | Cohort 5: Castrate-resistant Adenocarcinoma of the Prostate | Cohort 6: Castrate-resistant Adenocarcinoma of the Prostate | Cohort 7: Germline Mutated BRCA (gBRCAm) HER2- Adenocarcinoma of the Breast
Started | 1 | 4 | 5 | 11 | 5 | 11 | 1
Completed | 1 | 4 | 5 | 10 (11 participants were enrolled in cohort 4 and only 10 were included in the SA population.) | 5 | 10 (11 participants were enrolled in cohort 6 and only 10 were included in the SA population.) | 1
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — neither a de novo biopsy nor a research blood draw | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: NSCLC Monotherapy: Progressive disease on 1st line monotherapy anti-PD-1/-L1.
- Cohort 3: RCC With Clear Cell Component: Progressive disease on 2nd line monotherapy anti-PD-1/-L1; or progressive disease on 1st line combination of doublet anti-PD-1/-L1 with anti-CTLA-4; or progressive disease on 1st line combination of avelumab with axitinib or pembrolizumab with axitinib.
- Cohort 4: HR+ HER2- Adenocarcinoma of the Breast: Progressive disease on 1st line combination of doublet palbociclib with hormonal therapy.
- Cohort 7: gBRCAm HER2- Adenocarcinoma of the Breast: Progressive disease on a PARP inhibitor monotherapy in participants previously treated with chemotherapy in the neoadjuvant, adjuvant, or metastatic setting.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: NSCLC Monotherapy | Cohort 2: NSCLC Combination | Cohort 3: RCC With Clear Cell Component | Cohort 4: HR+ HER2- Adenocarcinoma of the Breast | Cohort 5: Castrate-resistant Adenocarcinoma of the Prostate | Cohort 6: Castrate-resistant Adenocarcinoma of the Prostate | Cohort 7: gBRCAm HER2- Adenocarcinoma of the Breast | Total
Number analyzed (Participants) | 1 | 4 | 5 | 10 | 5 | 10 | 1 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] — Data collected for Demographics and Baseline Characteristics Summary only in Safety Analysis Population
  Years | 73.0 | 70.8 (6.90) | 65.0 (9.11) | 66.6 (6.88) | 76.0 (9.85) | 64.7 (6.62) | 43.0 | 67.1 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants] — Data collected for Demographics and Baseline Characteristics Summary only in Safety Analysis Population
  Participants
    Female | 0 | 0 | 1 | 10 | 0 | 0 | 1 | 12
    Male | 1 | 4 | 4 | 0 | 5 | 10 | 0 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Data collected for Demographics and Baseline Characteristics Summary only in Safety Analysis Population
  Participants
    Hispanic or Latino | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 6
    Not Hispanic or Latino | 0 | 3 | 3 | 6 | 3 | 3 | 0 | 18
    Unknown or Not Reported | 0 | 1 | 1 | 1 | 1 | 7 | 1 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data collected for Demographics and Baseline Characteristics Summary only in Safety Analysis Population
  Participants
    White | 1 | 4 | 3 | 10 | 4 | 6 | 0 | 28
    Multiracial | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Not reported | 0 | 0 | 1 | 0 | 1 | 4 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in the Frequency of Gene Alterations Between Pre-treatment Tumor Samples (Archival) and Post-progression (De Novo) Tumor Biopsies
Description: Change in frequency is calculated by (frequency in de novo samples) - (frequency in archival samples). The frequency of each gene alteration is calculated as number of patients who harbored the alteration divided by the total number of patients in the cohort. Only gene alterations with variant allele frequency of 5% or greater were included in the analysis. Two different sequencing techniques were applied so 2 analysis sets were repeated for each cohort: targeted panel next-generation sequencing (NGS) and whole exome sequencing NGS.
Time Frame: Through study completion, approximately 3 months
Population: Number of Participants Analyzed shows the number of participants with available results for the corresponding gene alterations. Data for this outcome measure was not collected for Cohorts 1,2, 3 and 7 due to early termination of the study by Sponsor. Data for Cohorts 5 and 6 was combined to report combined results for Cohorts 5 and 6, to meet the sample size was deemed sufficient to generate informative summary statistics, as pre-specified in the Study Protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- HR+ HER2- Adenocarcinoma of the Breast With NGS Results: Participants in Cohort 4 with progressive disease on 1st line combination of doublet palbociclib with hormonal therapy and with NGS results from pre-treatment and post-progression tumor samples available.
- Castrate-resistant Adenocarcinoma of the Prostate With NGS Results: Participants in Cohort 5 & 6 with progressive disease on enzalutamide monotherapy and on abiraterone in combination with prednisone and with NGS results from pre-treatment and post-progression tumor samples available.
- HR+ HER2- Adenocarcinoma of the Breast With Whole Exome Sequencing NGS Results: Participants in Cohort 4 with progressive disease on 1st line combination of doublet palbociclib with hormonal therapy and with whole exome sequencing NGS results from pre-treatment and post-progression tumor samples available.
- Castrate-resistant Adenocarcinoma of the Prostate With Whole Exome Sequencing NGS Results: Participants in Cohort 5 & 6 with progressive disease on enzalutamide monotherapy and on abiraterone in combination with prednisone and with whole exome sequencing NGS results from pre-treatment and post-progression tumor samples available.
Arm/Group | HR+ HER2- Adenocarcinoma of the Breast With NGS Results | Castrate-resistant Adenocarcinoma of the Prostate With NGS Results | HR+ HER2- Adenocarcinoma of the Breast With Whole Exome Sequencing NGS Results | Castrate-resistant Adenocarcinoma of the Prostate With Whole Exome Sequencing NGS Results
Number analyzed (Participants) | 6 | 6 | 3 | 2
Percentage of Participants
  AKT1 c.238T>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  AKT1 c.238T>C | 16.7 [-28.9 to 56.4] |  |  |
  ARHGAP39 c.2000G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  ARHGAP39 c.2000G>A | 16.7 [-28.9 to 56.4] |  |  |
  ARHGAP39 c.2085G>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  ARHGAP39 c.2085G>C | -16.7 [-56.4 to 28.9] |  |  |
  ARID1A c.3145_3146dupCT: number analyzed (Participants) | 6 | 0 | 3 | 0
  ARID1A c.3145_3146dupCT | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  ARID1A c.3977dupC: number analyzed (Participants) | 6 | 0 | 0 | 0
  ARID1A c.3977dupC | 0.0 [-39.0 to 39.0] |  |  |
  ARID2 c.1803dupG: number analyzed (Participants) | 6 | 0 | 0 | 0
  ARID2 c.1803dupG | 0.0 [-39.0 to 39.0] |  |  |
  ASXL1 c.1934dupG: number analyzed (Participants) | 6 | 0 | 0 | 0
  ASXL1 c.1934dupG | 16.7 [-28.9 to 56.4] |  |  |
  ATM c.5557G>A: number analyzed (Participants) | 6 | 0 | 3 | 0
  ATM c.5557G>A | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  ATM c.5948A>G | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] | 0.0 [-65.8 to 65.8]
  AXIN1 c.1881G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  AXIN1 c.1881G>T | 16.7 [-28.9 to 56.4] |  |  |
  BAP1 c.179G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  BAP1 c.179G>A | 0.0 [-39.0 to 39.0] |  |  |
  BCLAF1 c.615_619delATCAGinsGTCAT: number analyzed (Participants) | 6 | 0 | 0 | 0
  BCLAF1 c.615_619delATCAGinsGTCAT | 16.7 [-28.9 to 56.4] |  |  |
  BCOR c.476C>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  BCOR c.476C>A | 16.7 [-28.9 to 56.4] |  |  |
  BRCA1 c.2612C>T: number analyzed (Participants) | 6 | 6 | 0 | 2
  BRCA1 c.2612C>T | 16.7 [-28.9 to 56.4] | 0.0 [-39.0 to 39.0] |  | 0.0 [-65.8 to 65.8]
  BRCA1 c.3113A>G: number analyzed (Participants) | 6 | 6 | 0 | 2
  BRCA1 c.3113A>G | 16.7 [-28.9 to 56.4] | 0.0 [-39.0 to 39.0] |  | 0.0 [-65.8 to 65.8]
  BRCA1 c.3548A>G: number analyzed (Participants) | 6 | 6 | 0 | 2
  BRCA1 c.3548A>G | 16.7 [-28.9 to 56.4] | 0.0 [-39.0 to 39.0] |  | 0.0 [-65.8 to 65.8]
  BRCA1 c.4837A>G: number analyzed (Participants) | 6 | 6 | 0 | 2
  BRCA1 c.4837A>G | 16.7 [-28.9 to 56.4] | 0.0 [-39.0 to 39.0] |  | 0.0 [-65.8 to 65.8]
  BRCA1 c.4956G>A: number analyzed (Participants) | 6 | 6 | 0 | 0
  BRCA1 c.4956G>A | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] |  |
  BRCA2 c.1114A>C: number analyzed (Participants) | 6 | 6 | 3 | 0
  BRCA2 c.1114A>C | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] |
  BRCA2 c.2803G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  BRCA2 c.2803G>A | 0.0 [-39.0 to 39.0] |  |  |
  BRCA2 c.7397T>C | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] | 0.0 [-65.8 to 65.8]
  BRCA2 c.9976A>T: number analyzed (Participants) | 6 | 0 | 3 | 0
  BRCA2 c.9976A>T | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  BRIP1 c.14G>C: number analyzed (Participants) | 6 | 0 | 3 | 0
  BRIP1 c.14G>C | -16.7 [-56.4 to 28.9] |  | -33.3 [-79.2 to 41.5] |
  BRIP1 c.2755T>C | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] | 0.0 [-65.8 to 65.8]
  CBR3 c.730G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  CBR3 c.730G>A | 16.7 [-28.9 to 56.4] |  |  |
  CCNE1 c.1117G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  CCNE1 c.1117G>A | -16.7 [-56.4 to 28.9] |  |  |
  CD22 c.757G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  CD22 c.757G>T | -16.7 [-56.4 to 28.9] |  |  |
  CD3EAP c.1516C>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  CD3EAP c.1516C>A | 16.7 [-28.9 to 56.4] |  |  |
  CDH1 c.1269delT: number analyzed (Participants) | 6 | 0 | 0 | 0
  CDH1 c.1269delT | 0.0 [-39.0 to 39.0] |  |  |
  CDH1 c.466T>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  CDH1 c.466T>A | 0.0 [-39.0 to 39.0] |  |  |
  CREBBP c.1792C>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  CREBBP c.1792C>T | 16.7 [-28.9 to 56.4] |  |  |
  CSF3R c.14G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  CSF3R c.14G>T | 0.0 [-39.0 to 39.0] |  |  |
  DNM2 c.1782-5delC: number analyzed (Participants) | 6 | 0 | 0 | 0
  DNM2 c.1782-5delC | 0.0 [-39.0 to 39.0] |  |  |
  DPYD c.1471G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  DPYD c.1471G>T | 16.7 [-28.9 to 56.4] |  |  |
  DYNC2H1 c.1714A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  DYNC2H1 c.1714A>G | -16.7 [-56.4 to 28.9] |  |  |
  ECH1 c.122A>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  ECH1 c.122A>C | 16.7 [-28.9 to 56.4] |  |  |
  ERBB2 c.1958C>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  ERBB2 c.1958C>G | 16.7 [-28.9 to 56.4] |  |  |
  ERBB2 c.2446C>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  ERBB2 c.2446C>T | -16.7 [-56.4 to 28.9] |  |  |
  ERCC5 c.440C>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  ERCC5 c.440C>G | -16.7 [-56.4 to 28.9] |  |  |
  ESR1 c.1609T>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  ESR1 c.1609T>A | 16.7 [-28.9 to 56.4] |  |  |
  ESR1 c.1610_1613delATGAinsGTGG: number analyzed (Participants) | 6 | 0 | 0 | 0
  ESR1 c.1610_1613delATGAinsGTGG | 16.7 [-28.9 to 56.4] |  |  |
  ESR1 c.1613A>G: number analyzed (Participants) | 6 | 0 | 3 | 0
  ESR1 c.1613A>G | 16.7 [-28.9 to 56.4] |  | 33.3 [-41.5 to 79.2] |
  FAM175A c.826_828delGAG: number analyzed (Participants) | 6 | 0 | 0 | 0
  FAM175A c.826_828delGAG | -16.7 [-56.4 to 28.9] |  |  |
  FANCA c.2426G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  FANCA c.2426G>A | 16.7 [-28.9 to 56.4] |  |  |
  FANCD2 c.1214A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  FANCD2 c.1214A>G | -16.7 [-56.4 to 28.9] |  |  |
  FANCE c.17C>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  FANCE c.17C>G | -16.7 [-16.7 to 28.9] |  |  |
  FAT1 c.3818A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  FAT1 c.3818A>G | 16.7 [-28.9 to 56.4] |  |  |
  FGF9 c.375T>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  FGF9 c.375T>A | 0.0 [-39.0 to 39.0] |  |  |
  FGFR1 c.358+4G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  FGFR1 c.358+4G>A | -16.7 [-56.4 to 28.9] |  |  |
  FGFR1OP c.985-6_985-5dupTT: number analyzed (Participants) | 6 | 0 | 0 | 0
  FGFR1OP c.985-6_985-5dupTT | -16.7 [-56.4 to 28.9] |  |  |
  FLT4 c.1019G>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  FLT4 c.1019G>C | 16.7 [-28.9 to 56.4] |  |  |
  FOXA1 c.247G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  FOXA1 c.247G>A | 16.7 [-28.9 to 56.4] |  |  |
  FOXA1 c.801G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  FOXA1 c.801G>T | 0.0 [-39.0 to 39.0] |  |  |
  FOXA1 c.874G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  FOXA1 c.874G>T | 16.7 [-28.9 to 56.4] |  |  |
  FOXQ1 c.1013A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  FOXQ1 c.1013A>G | -16.7 [-56.4 to 28.9] |  |  |
  FOXQ1 c.895G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  FOXQ1 c.895G>A | 16.7 [-28.9 to 56.4] |  |  |
  FRS2 c.236G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  FRS2 c.236G>T | 16.7 [-28.9 to 56.4] |  |  |
  GATA2 c.527C>T: number analyzed (Participants) | 6 | 0 | 3 | 0
  GATA2 c.527C>T | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  GATA3 c.1223_1224insA: number analyzed (Participants) | 6 | 0 | 3 | 0
  GATA3 c.1223_1224insA | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  GNAS c.521G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  GNAS c.521G>A | 16.7 [-28.9 to 56.4] |  |  |
  GOT2 c.1037T>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  GOT2 c.1037T>G | 16.7 [-28.9 to 56.4] |  |  |
  HEATR1 c.6347-4_6347-3dupTT: number analyzed (Participants) | 6 | 0 | 0 | 0
  HEATR1 c.6347-4_6347-3dupTT | -16.7 [-56.4 to 28.9] |  |  |
  IRF2 c.744G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  IRF2 c.744G>A | 16.7 [-28.9 to 56.4] |  |  |
  IRS2 c.3170G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  IRS2 c.3170G>A | 16.7 [-28.9 to 56.4] |  |  |
  ITPKB c.1222T>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  ITPKB c.1222T>G | 16.7 [-28.9 to 56.4] |  |  |
  JAK1 c.1252G>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  JAK1 c.1252G>C | 16.7 [-28.9 to 56.4] |  |  |
  JAK2 c.2743G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  JAK2 c.2743G>T | 16.7 [-28.9 to 56.4] |  |  |
  JAK3 c.757A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  JAK3 c.757A>G | 16.7 [-28.9 to 56.4] |  |  |
  KDM6A c.2859-5delT: number analyzed (Participants) | 6 | 6 | 0 | 0
  KDM6A c.2859-5delT | -16.7 [-56.4 to 28.9] | 16.7 [-28.9 to 56.4] |  |
  KDR c.2921G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  KDR c.2921G>T | -16.7 [-56.4 to 28.9] |  |  |
  KMT2C c.2536delG: number analyzed (Participants) | 6 | 0 | 3 | 0
  KMT2C c.2536delG | 0.0 [-39.0 to 39.0] |  | 0 [-56.1 to 56.1] |
  KMT2C c.4270C>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  KMT2C c.4270C>T | 16.7 [-28.9 to 56.4] |  |  |
  LMAN1 c.823-2dupA: number analyzed (Participants) | 6 | 0 | 0 | 0
  LMAN1 c.823-2dupA | -16.7 [-56.4 to 28.9] |  |  |
  LRP1B c.143A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  LRP1B c.143A>G | 16.7 [-28.9 to 56.4] |  |  |
  LRP1B c.5737G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  LRP1B c.5737G>A | -16.7 [-56.4 to 28.9] |  |  |
  LTN1 c.1717A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  LTN1 c.1717A>G | 16.7 [-28.9 to 56.4] |  |  |
  LYN c.475G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  LYN c.475G>T | 16.7 [-28.9 to 56.4] |  |  |
  MAP2K4 c.179C>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  MAP2K4 c.179C>A | -16.7 [-56.4 to 28.9] |  |  |
  MED12 c.1364G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  MED12 c.1364G>T | 16.7 [-28.9 to 56.4] |  |  |
  MGMT c.520A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  MGMT c.520A>G | 16.7 [-28.9 to 56.4] |  |  |
  MGMT c.626A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  MGMT c.626A>G | 16.7 [-28.9 to 56.4] |  |  |
  MLH1 c.655A>G: number analyzed (Participants) | 6 | 6 | 3 | 0
  MLH1 c.655A>G | 16.7 [-28.9 to 56.4] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] |
  MSH2 c.1748A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  MSH2 c.1748A>G | 0.0 [-39.0 to 39.0] |  |  |
  MSH6 c.116G>A | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] | 0.0 [-65.8 to 65.8]
  MSH6 c.3557-4dupT: number analyzed (Participants) | 6 | 0 | 0 | 0
  MSH6 c.3557-4dupT | 16.7 [-28.9 to 56.4] |  |  |
  MTHFR c.1286A>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  MTHFR c.1286A>C | 16.7 [-28.9 to 56.4] |  |  |
  MUTYH c.1014G>C: number analyzed (Participants) | 6 | 6 | 3 | 0
  MUTYH c.1014G>C | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] |
  MUTYH c.1187G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  MUTYH c.1187G>A | 0.0 [-39.0 to 39.0] |  |  |
  MYB c.1781C>G: number analyzed (Participants) | 6 | 0 | 3 | 0
  MYB c.1781C>G | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  NBN c.553G>C | 0.0 [-39.0 to 39.0] | -33.3 [-70.0 to 18.7] | 0.0 [-56.1 to 56.1] | 0.0 [-65.8 to 65.8]
  NBN c.683T>G: number analyzed (Participants) | 6 | 0 | 3 | 0
  NBN c.683T>G | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  NCOR1 c.4135G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  NCOR1 c.4135G>T | 0.0 [-39.0 to 39.0] |  |  |
  NCOR2 c.1597G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  NCOR2 c.1597G>A | 0.0 [-39.0 to 39.0] |  |  |
  NF1 c.7063-1G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  NF1 c.7063-1G>T | -16.7 [-56.4 to 28.9] |  |  |
  NF1 c.849T>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  NF1 c.849T>G | 16.7 [-28.9 to 56.4] |  |  |
  NOTCH1 c.2588-4G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  NOTCH1 c.2588-4G>A | 16.7 [-28.9 to 56.4] |  |  |
  NOTCH2 c.3522+3G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  NOTCH2 c.3522+3G>A | 16.7 [-28.9 to 56.4] |  |  |
  NOTCH3 c.539C>T: number analyzed (Participants) | 6 | 0 | 3 | 0
  NOTCH3 c.539C>T | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  NTRK1 c.1806-4delA: number analyzed (Participants) | 6 | 0 | 0 | 0
  NTRK1 c.1806-4delA | 16.7 [-28.9 to 56.4] |  |  |
  NUP98 c.3310G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  NUP98 c.3310G>A | 16.7 [-28.9 to 56.4] |  |  |
  PALB2 c.1676A>G | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] | 0.0 [-65.8 to 65.8]
  PALB2 c.2014G>C | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] | 0.0 [-65.8 to 65.8]
  PIK3CA c.1035T>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  PIK3CA c.1035T>A | 0.0 [-39.0 to 39.0] |  |  |
  PIK3CA c.1633G>A: number analyzed (Participants) | 6 | 0 | 3 | 0
  PIK3CA c.1633G>A | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  PIK3CA c.3140A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  PIK3CA c.3140A>G | 0.0 [-39.0 to 39.0] |  |  |
  PIK3CG c.41A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  PIK3CG c.41A>G | -16.7 [-56.4 to 28.9] |  |  |
  PLCG2 c.2011A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  PLCG2 c.2011A>G | 16.7 [-28.9 to 56.4] |  |  |
  PMS2 c.13G>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  PMS2 c.13G>C | 0.0 [-39.0 to 39.0] |  |  |
  PMS2 c.1408C>T: number analyzed (Participants) | 6 | 6 | 3 | 0
  PMS2 c.1408C>T | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] |
  PMS2 c.1454C>A: number analyzed (Participants) | 6 | 0 | 3 | 0
  PMS2 c.1454C>A | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  PMS2 c.1621A>G | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] | 0.0 [-65.8 to 65.8]
  PMS2 c.2570G>C | 0.0 [-39.0 to 39.0] | 33.3 [-18.7 to 70.0] | 0.0 [-56.1 to 56.1] | 50.0 [-48.6 to 90.5]
  PMS2 c.89A>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  PMS2 c.89A>G | 0.0 [-39.0 to 39.0] |  |  |
  POLD1 c.2959delG: number analyzed (Participants) | 6 | 0 | 0 | 0
  POLD1 c.2959delG | -16.7 [-56.4 to 28.9] |  |  |
  PRKDC c.6424C>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  PRKDC c.6424C>T | -16.7 [-56.4 to 28.9] |  |  |
  PTCH1 c.3746C>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  PTCH1 c.3746C>T | 16.7 [-28.9 to 56.4] |  |  |
  PTCH2 c.2134G>A: number analyzed (Participants) | 6 | 0 | 3 | 0
  PTCH2 c.2134G>A | 0.0 [-39.0 to 39.0] |  | 0 [-56.1 to 56.1] |
  PTPN13 c.4097T>A: number analyzed (Participants) | 6 | 0 | 3 | 0
  PTPN13 c.4097T>A | -16.7 [-56.4 to 28.9] |  | -33.3 [-79.2 to 41.5] |
  PTPN13 c.5683A>T: number analyzed (Participants) | 6 | 0 | 3 | 0
  PTPN13 c.5683A>T | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  PTPN13 c.6256T>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  PTPN13 c.6256T>G | 16.7 [-28.9 to 56.4] |  |  |
  PUS3 c.1380G>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  PUS3 c.1380G>C | 16.7 [-28.9 to 56.4] |  |  |
  RAD51C c.376G>A: number analyzed (Participants) | 6 | 6 | 3 | 0
  RAD51C c.376G>A | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] |
  RAD51D c.494G>A: number analyzed (Participants) | 6 | 0 | 3 | 0
  RAD51D c.494G>A | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  RIT1 c.625G>C: number analyzed (Participants) | 6 | 0 | 3 | 0
  RIT1 c.625G>C | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  RNF43 c.1252C>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  RNF43 c.1252C>A | 16.7 [-28.9 to 56.4] |  |  |
  ROS1 c.1775_1777delGTG: number analyzed (Participants) | 6 | 0 | 3 | 0
  ROS1 c.1775_1777delGTG | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  RSF1 c.3025G>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  RSF1 c.3025G>C | -16.7 [-56.4 to 28.9] |  |  |
  SF3B1 c.2077+4A>G: number analyzed (Participants) | 6 | 0 | 3 | 0
  SF3B1 c.2077+4A>G | 16.7 [-28.9 to 56.4] |  | 33.3 [-41.5 to 79.2] |
  SOD2 c.47T>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  SOD2 c.47T>C | 16.7 [-28.9 to 56.4] |  |  |
  SYNE1 c.18758G>A: number analyzed (Participants) | 6 | 0 | 3 | 0
  SYNE1 c.18758G>A | 16.7 [-28.9 to 56.4] |  | 33.3 [-41.5 to 79.2] |
  TBC1D12 c.1246C>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  TBC1D12 c.1246C>T | -16.7 [-56.4 to 28.9] |  |  |
  TBC1D9B c.3356A>C: number analyzed (Participants) | 6 | 0 | 0 | 0
  TBC1D9B c.3356A>C | 16.7 [-28.9 to 56.4] |  |  |
  TBX3 c.364G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  TBX3 c.364G>A | 0.0 [-39.0 to 39.0] |  |  |
  TBX3 c.820_827dupCCCGAAAC: number analyzed (Participants) | 6 | 0 | 0 | 0
  TBX3 c.820_827dupCCCGAAAC | 0.0 [-39.0 to 39.0] |  |  |
  TCF3 c.737C>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  TCF3 c.737C>T | -16.7 [-56.4 to 28.9] |  |  |
  TERT c.215G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  TERT c.215G>A | 16.7 [-28.9 to 56.4] |  |  |
  TGFBR2 c.530-4T>A: number analyzed (Participants) | 6 | 6 | 0 | 0
  TGFBR2 c.530-4T>A | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] |  |
  TP53 c.215C>G | 0.0 [-39.0 to 39.0] | 0.0 [-39.0 to 39.0] | 0.0 [-56.1 to 56.1] | 0.0 [-65.8 to 65.8]
  TP53 c.388delC: number analyzed (Participants) | 6 | 0 | 3 | 0
  TP53 c.388delC | 0.0 [-39.0 to 39.0] |  | 0.0 [-56.1 to 56.1] |
  TP53 c.782+1G>A: number analyzed (Participants) | 6 | 0 | 0 | 0
  TP53 c.782+1G>A | 0.0 [-39.0 to 39.0] |  |  |
  TUSC3 c.99_101delGCT: number analyzed (Participants) | 6 | 0 | 0 | 0
  TUSC3 c.99_101delGCT | -16.7 [-56.4 to 28.9] |  |  |
  ZFHX3 c.10931G>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  ZFHX3 c.10931G>T | -16.7 [-56.4 to 28.9] |  |  |
  ZFHX3 c.1135C>G: number analyzed (Participants) | 6 | 0 | 0 | 0
  ZFHX3 c.1135C>G | 16.7 [-28.9 to 56.4] |  |  |
  ZFHX3 c.1631C>T: number analyzed (Participants) | 6 | 0 | 0 | 0
  ZFHX3 c.1631C>T | -16.7 [-56.4 to 28.9] |  |  |
  ZFHX3 c.2833T>G: number analyzed (Participants) | 6 | 0 | 3 | 0
  ZFHX3 c.2833T>G | -16.7 [-56.4 to 28.9] |  | -33.3 [-79.2 to 41.5] |
  ALK c.1043C>A: number analyzed (Participants) | 0 | 6 | 0 | 0
  ALK c.1043C>A |  | 16.7 [-28.9 to 56.4] |  |
  APLNR c.349G>A: number analyzed (Participants) | 0 | 6 | 0 | 0
  APLNR c.349G>A |  | 0.0 [-39.0 to 39.0] |  |
  CARD11 c.988G>A: number analyzed (Participants) | 0 | 6 | 0 | 0
  CARD11 c.988G>A |  | 0.0 [-39.0 to 39.0] |  |
  CHD4 c.4060G>C: number analyzed (Participants) | 0 | 6 | 0 | 2
  CHD4 c.4060G>C |  | -16.7 [-56.4 to 28.9] |  | 0.0 [-65.8 to 65.8]
  EGFR c.1008G>A: number analyzed (Participants) | 0 | 6 | 0 | 2
  EGFR c.1008G>A |  | 0.0 [-39.0 to 39.0] |  | 0.0 [-65.8 to 65.8]
  EP300 c.6613A>C: number analyzed (Participants) | 0 | 6 | 0 | 0
  EP300 c.6613A>C |  | -16.7 [-56.4 to 28.9] |  |
  ERCC6 c.3661C>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  ERCC6 c.3661C>T |  | -16.7 [-56.4 to 28.9] |  |
  ERG c.1455_1461delCTACTAA: number analyzed (Participants) | 0 | 6 | 0 | 0
  ERG c.1455_1461delCTACTAA |  | -16.7 [-56.4 to 28.9] |  |
  EZH2 c.848C>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  EZH2 c.848C>T |  | 0.0 [-39.0 to 39.0] |  |
  FBXO11 c.164_169delAGCAGC: number analyzed (Participants) | 0 | 6 | 0 | 0
  FBXO11 c.164_169delAGCAGC |  | 16.7 [-28.9 to 56.4] |  |
  FLT4 c.2405G>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  FLT4 c.2405G>T |  | -16.7 [-56.4 to 28.9] |  |
  FOXO1 c.302C>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  FOXO1 c.302C>T |  | 16.7 [-28.9 to 56.4] |  |
  GNAQ c.303C>A: number analyzed (Participants) | 0 | 6 | 0 | 0
  GNAQ c.303C>A |  | -16.7 [-56.4 to 28.9] |  |
  HOTS c.233_236delTACTinsCACC: number analyzed (Participants) | 0 | 6 | 0 | 0
  HOTS c.233_236delTACTinsCACC |  | 16.7 [-28.9 to 56.4] |  |
  IRS2 c.1242C>A: number analyzed (Participants) | 0 | 6 | 0 | 0
  IRS2 c.1242C>A |  | -16.7 [-56.4 to 28.9] |  |
  KDM5C c.3019C>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  KDM5C c.3019C>T |  | -16.7 [-56.4 to 28.9] |  |
  KIT c.597delA: number analyzed (Participants) | 0 | 6 | 0 | 0
  KIT c.597delA |  | -16.7 [-56.4 to 28.9] |  |
  KMT2A c.9400C>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  KMT2A c.9400C>T |  | 16.7 [-28.9 to 56.4] |  |
  KMT2B c.26G>A: number analyzed (Participants) | 0 | 6 | 0 | 0
  KMT2B c.26G>A |  | -16.7 [-56.4 to 28.9] |  |
  KMT2C c.4845G>A: number analyzed (Participants) | 0 | 6 | 0 | 2
  KMT2C c.4845G>A |  | 16.7 [-28.9 to 56.4] |  | 50.0 [-48.6 to 90.5]
  LRP1B c.4439G>A: number analyzed (Participants) | 0 | 6 | 0 | 0
  LRP1B c.4439G>A |  | 0.0 [-39.0 to 39.0] |  |
  MAGEA10 c.1021G>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  MAGEA10 c.1021G>T |  | -16.7 [-56.4 to 28.9] |  |
  MAP3K1 c.4292A>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  MAP3K1 c.4292A>T |  | 0.0 [-39.0 to 39.0] |  |
  MET c.2318C>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  MET c.2318C>T |  | 0.0 [-39.0 to 39.0] |  |
  MSH6 c.1186C>G: number analyzed (Participants) | 0 | 6 | 0 | 0
  MSH6 c.1186C>G |  | 0.0 [-39.0 to 39.0] |  |
  MSH6 c.1486T>G: number analyzed (Participants) | 0 | 6 | 0 | 0
  MSH6 c.1486T>G |  | 0.0 [-39.0 to 39.0] |  |
  MUTYH c.64G>A: number analyzed (Participants) | 0 | 6 | 0 | 2
  MUTYH c.64G>A |  | 0.0 [-39.0 to 39.0] |  | 0.0 [-65.8 to 65.8]
  MYH11 c.5819dupC: number analyzed (Participants) | 0 | 6 | 0 | 0
  MYH11 c.5819dupC |  | 16.7 [-28.9 to 56.4] |  |
  NF1 c.1082G>C: number analyzed (Participants) | 0 | 6 | 0 | 0
  NF1 c.1082G>C |  | 0.0 [-39.0 to 39.0] |  |
  NOTCH2 c.17_18delCC: number analyzed (Participants) | 0 | 6 | 0 | 0
  NOTCH2 c.17_18delCC |  | -16.7 [-56.4 to 28.9] |  |
  NTRK3 c.137G>C: number analyzed (Participants) | 0 | 6 | 0 | 0
  NTRK3 c.137G>C |  | 16.7 [-28.9 to 56.4] |  |
  PALB2 c.2993G>A: number analyzed (Participants) | 0 | 6 | 0 | 2
  PALB2 c.2993G>A |  | 0.0 [-39.0 to 39.0] |  | 0.0 [-65.8 to 65.8]
  PALLD c.270_275dupCCCGCC: number analyzed (Participants) | 0 | 6 | 0 | 0
  PALLD c.270_275dupCCCGCC |  | -16.7 [-56.4 to 28.9] |  |
  PAX8 c.352G>A: number analyzed (Participants) | 0 | 6 | 0 | 0
  PAX8 c.352G>A |  | -16.7 [-56.4 to 28.9] |  |
  PDGFRB c.1543G>C: number analyzed (Participants) | 0 | 6 | 0 | 2
  PDGFRB c.1543G>C |  | -16.7 [-56.4 to 28.9] |  | -50.0 [-90.5 to 48.6]
  PIK3R1 c.1690A>G: number analyzed (Participants) | 0 | 6 | 0 | 0
  PIK3R1 c.1690A>G |  | 16.7 [-28.9 to 56.4] |  |
  PIK3R1 c.935delC: number analyzed (Participants) | 0 | 6 | 0 | 0
  PIK3R1 c.935delC |  | -16.7 [-56.4 to 28.9] |  |
  PIK3R2 c.2047T>G: number analyzed (Participants) | 0 | 6 | 0 | 2
  PIK3R2 c.2047T>G |  | 16.7 [-28.9 to 56.4] |  | 0.0 [-65.8 to 65.8]
  PLCG1 c.1825C>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  PLCG1 c.1825C>T |  | 16.7 [-28.9 to 56.4] |  |
  PLCG2 c.2114G>A: number analyzed (Participants) | 0 | 6 | 0 | 2
  PLCG2 c.2114G>A |  | 0.0 [-39.0 to 39.0] |  | 0.0 [-65.8 to 65.8]
  PMS2 c.1789A>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  PMS2 c.1789A>T |  | 0.0 [-39.0 to 39.0] |  |
  PMS2 c.706-4delT: number analyzed (Participants) | 0 | 6 | 0 | 0
  PMS2 c.706-4delT |  | 16.7 [-28.9 to 56.4] |  |
  PTEN c.900delC: number analyzed (Participants) | 0 | 6 | 0 | 0
  PTEN c.900delC |  | -16.7 [-56.4 to 28.9] |  |
  PTPRD c.2069A>G: number analyzed (Participants) | 0 | 6 | 0 | 0
  PTPRD c.2069A>G |  | 0.0 [-39.0 to 39.0] |  |
  RB1 c.1466G>A: number analyzed (Participants) | 0 | 6 | 0 | 2
  RB1 c.1466G>A |  | 16.7 [-28.9 to 56.4] |  | 50.0 [-48.6 to 90.5]
  RNF139 c.135C>G: number analyzed (Participants) | 0 | 6 | 0 | 0
  RNF139 c.135C>G |  | -16.7 [-56.4 to 28.9] |  |
  ROS1 c.3416A>G: number analyzed (Participants) | 0 | 6 | 0 | 2
  ROS1 c.3416A>G |  | 16.7 [-28.9 to 56.4] |  | 50.0 [-48.6 to 90.5]
  SPOP c.260A>G: number analyzed (Participants) | 0 | 6 | 0 | 0
  SPOP c.260A>G |  | 0.0 [-39.0 to 39.0] |  |
  SYNE1 c.25403G>A: number analyzed (Participants) | 0 | 6 | 0 | 0
  SYNE1 c.25403G>A |  | 0.0 [-39.0 to 39.0] |  |
  TCF3 c.1643G>A: number analyzed (Participants) | 0 | 6 | 0 | 0
  TCF3 c.1643G>A |  | -16.7 [-56.4 to 28.9] |  |
  TEP1 c.3649C>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  TEP1 c.3649C>T |  | 0.0 [-39.0 to 39.0] |  |
  TP53 c.993G>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  TP53 c.993G>T |  | -16.7 [-56.4 to 28.9] |  |
  TP53 c.994-2A>G: number analyzed (Participants) | 0 | 6 | 0 | 0
  TP53 c.994-2A>G |  | 16.7 [-28.9 to 56.4] |  |
  U2AF1 c.101C>T: number analyzed (Participants) | 0 | 6 | 0 | 0
  U2AF1 c.101C>T |  | -16.7 [-56.4 to 28.9] |  |
  ZFHX3 c.11065A>G: number analyzed (Participants) | 0 | 6 | 0 | 0
  ZFHX3 c.11065A>G |  | 16.7 [-28.9 to 56.4] |  |
  AATK c.65C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  AATK c.65C>T |  |  | -33.3 [-79.2 to 41.5] |
  ABCC9 c.4535C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ABCC9 c.4535C>T |  |  | 0.0 [-56.1 to 56.1] |
  ACADS c.989G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ACADS c.989G>A |  |  | 33.3 [-41.5 to 79.2] |
  ACAP3 c.1990C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ACAP3 c.1990C>T |  |  | -33.3 [-79.2 to 41.5] |
  ACSL4 c.106G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ACSL4 c.106G>A |  |  | -33.3 [-79.2 to 41.5] |
  ADAMTS13 c.3287G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ADAMTS13 c.3287G>A |  |  | 33.3 [-41.5 to 79.2] |
  ADAMTS7 c.227G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ADAMTS7 c.227G>A |  |  | 33.3 [-41.5 to 79.2] |
  ADCY5 c.778C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ADCY5 c.778C>T |  |  | -33.3 [-79.2 to 41.5] |
  ADGRE2 c.934C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ADGRE2 c.934C>A |  |  | 33.3 [-41.5 to 79.2] |
  ADGRE3 c.1411G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ADGRE3 c.1411G>A |  |  | -33.3 [-79.2 to 41.5] |
  ADGRF2 c.680C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ADGRF2 c.680C>T |  |  | -33.3 [-79.2 to 41.5] |
  ADGRG3 c.1394C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ADGRG3 c.1394C>T |  |  | -33.3 [-79.2 to 41.5] |
  ADH4 c.1174delA: number analyzed (Participants) | 0 | 0 | 3 | 0
  ADH4 c.1174delA |  |  | -33.3 [-79.2 to 41.5] |
  AEBP1 c.799G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  AEBP1 c.799G>A |  |  | -33.3 [-79.2 to 41.5] |
  AGFG2 c.340C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  AGFG2 c.340C>A |  |  | 33.3 [-41.5 to 79.2] |
  AGPAT4 c.853C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  AGPAT4 c.853C>T |  |  | 0.0 [-56.1 to 56.1] |
  AGRN c.184C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  AGRN c.184C>A |  |  | 33.3 [-41.5 to 79.2] |
  AGRN c.3157G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  AGRN c.3157G>C |  |  | 0.0 [-56.1 to 56.1] |
  AHNAK2 c.13479G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  AHNAK2 c.13479G>A |  |  | -33.3 [-79.2 to 41.5] |
  AHNAK2 c.9650T>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  AHNAK2 c.9650T>C |  |  | -33.3 [-79.2 to 41.5] |
  AKNA c.3907T>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  AKNA c.3907T>C |  |  | 33.3 [-41.5 to 79.2] |
  ALS2CL c.14A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  ALS2CL c.14A>G |  |  | -33.3 [-79.2 to 41.5] |
  ANKRD61 c.323C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  ANKRD61 c.323C>G |  |  | 33.3 [-41.5 to 79.2] |
  ANKS1A c.157_159delGGC: number analyzed (Participants) | 0 | 0 | 3 | 0
  ANKS1A c.157_159delGGC |  |  | -33.3 [-79.2 to 41.5] |
  ANKS1B c.2548C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ANKS1B c.2548C>A |  |  | -33.3 [-79.2 to 41.5] |
  ANTXR1 c.1121A>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  ANTXR1 c.1121A>C |  |  | 33.3 [-41.5 to 79.2] |
  ANTXR2 c.940G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ANTXR2 c.940G>A |  |  | -33.3 [-79.2 to 41.5] |
  APC2 c.1312C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  APC2 c.1312C>T |  |  | -33.3 [-79.2 to 41.5] |
  APLP1 c.1243C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  APLP1 c.1243C>T |  |  | 0.0 [-56.1 to 56.1] |
  ARF6 c.352_354delCTC: number analyzed (Participants) | 0 | 0 | 3 | 0
  ARF6 c.352_354delCTC |  |  | 33.3 [-41.5 to 79.2] |
  ARHGAP6 c.1585G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  ARHGAP6 c.1585G>C |  |  | 33.3 [-41.5 to 79.2] |
  ARHGEF1 c.2031_2033delGCT: number analyzed (Participants) | 0 | 0 | 3 | 0
  ARHGEF1 c.2031_2033delGCT |  |  | 33.3 [-41.5 to 79.2] |
  ARHGEF19 c.1379C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ARHGEF19 c.1379C>T |  |  | 33.3 [-41.5 to 79.2] |
  ARHGEF7 c.2072G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ARHGEF7 c.2072G>A |  |  | -33.3 [-79.2 to 41.5] |
  ARL10 c.53C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ARL10 c.53C>T |  |  | 33.3 [-41.5 to 79.2] |
  ARL6IP4 c.902_904delAGA: number analyzed (Participants) | 0 | 0 | 3 | 0
  ARL6IP4 c.902_904delAGA |  |  | -33.3 [-79.2 to 41.5] |
  ARRDC4 c.227C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ARRDC4 c.227C>T |  |  | -33.3 [-79.2 to 41.5] |
  ARSI c.312G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ARSI c.312G>A |  |  | -33.3 [-79.2 to 41.5] |
  ASCC3 c.5962A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  ASCC3 c.5962A>G |  |  | 0.0 [-56.1 to 56.1] |
  ASH1L c.8522G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ASH1L c.8522G>A |  |  | -33.3 [-79.2 to 41.5] |
  ASPRV1 c.985G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ASPRV1 c.985G>T |  |  | 33.3 [-41.5 to 79.2] |
  ATM c.3403-4dupT: number analyzed (Participants) | 0 | 0 | 3 | 2
  ATM c.3403-4dupT |  |  | 0.0 [-56.1 to 56.1] | 0.0 [-65.8 to 65.8]
  ATP13A2 c.2984C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ATP13A2 c.2984C>T |  |  | -33.3 [-79.2 to 41.5] |
  ATP2C2 c.2192delA: number analyzed (Participants) | 0 | 0 | 3 | 0
  ATP2C2 c.2192delA |  |  | 33.3 [-41.5 to 79.2] |
  ATP6AP1 c.508A>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  ATP6AP1 c.508A>C |  |  | -33.3 [-79.2 to 41.5] |
  ATP7A c.3388C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ATP7A c.3388C>A |  |  | -33.3 [-79.2 to 41.5] |
  ATRN c.263_268delCGGCGG: number analyzed (Participants) | 0 | 0 | 3 | 0
  ATRN c.263_268delCGGCGG |  |  | 33.3 [-41.5 to 79.2] |
  B3GLCT c.517G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  B3GLCT c.517G>A |  |  | -33.3 [-79.2 to 41.5] |
  B4GALNT2 c.1414G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  B4GALNT2 c.1414G>A |  |  | 33.3 [-41.5 to 79.2] |
  B4GALT7 c.431T>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  B4GALT7 c.431T>C |  |  | 33.3 [-41.5 to 79.2] |
  BEGAIN c.1231G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  BEGAIN c.1231G>A |  |  | -33.3 [-79.2 to 41.5] |
  BEST1 c.273C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  BEST1 c.273C>G |  |  | -33.3 [-79.2 to 41.5] |
  BET1 c.327dupT: number analyzed (Participants) | 0 | 0 | 3 | 0
  BET1 c.327dupT |  |  | -33.3 [-79.2 to 41.5] |
  BNC1 c.86G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  BNC1 c.86G>A |  |  | -33.3 [-79.2 to 41.5] |
  BOC c.896G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  BOC c.896G>A |  |  | -33.3 [-79.2 to 41.5] |
  BPIFB4 c.1146G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  BPIFB4 c.1146G>A |  |  | -33.3 [-79.2 to 41.5] |
  BRPF1 c.3069C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  BRPF1 c.3069C>T |  |  | -33.3 [-79.2 to 41.5] |
  BRPF1 c.823G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  BRPF1 c.823G>C |  |  | 0.0 [-56.1 to 56.1] |
  BRWD3 c.3188G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  BRWD3 c.3188G>T |  |  | -33.3 [-79.2 to 41.5] |
  BTBD17 c.106G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  BTBD17 c.106G>A |  |  | -33.3 [-79.2 to 41.5] |
  C10orf88 c.401dupA: number analyzed (Participants) | 0 | 0 | 3 | 0
  C10orf88 c.401dupA |  |  | -33.3 [-79.2 to 41.5] |
  C16orf47 c.329G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  C16orf47 c.329G>A |  |  | -33.3 [-79.2 to 41.5] |
  C16orf95 c.407G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  C16orf95 c.407G>A |  |  | -33.3 [-79.2 to 41.5] |
  C17orf100 c.71C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  C17orf100 c.71C>T |  |  | -33.3 [-79.2 to 41.5] |
  C17orf105 c.97G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  C17orf105 c.97G>A |  |  | 33.3 [-41.5 to 79.2] |
  C1QL4 c.185G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  C1QL4 c.185G>A |  |  | -33.3 [-79.2 to 41.5] |
  C1orf122 c.17G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  C1orf122 c.17G>A |  |  | -33.3 [-79.2 to 41.5] |
  C1orf168 c.2134G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  C1orf168 c.2134G>A |  |  | -33.3 [-79.2 to 41.5] |
  C3 c.3566_3567delTG: number analyzed (Participants) | 0 | 0 | 3 | 0
  C3 c.3566_3567delTG |  |  | 33.3 [-41.5 to 79.2] |
  C5orf60 c.770G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  C5orf60 c.770G>A |  |  | -33.3 [-79.2 to 41.5] |
  C7orf31 c.931A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  C7orf31 c.931A>G |  |  | 0.0 [-56.1 to 56.1] |
  CACNA1C c.169G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CACNA1C c.169G>A |  |  | -33.3 [-79.2 to 41.5] |
  CACNA1D c.26_28delAAA: number analyzed (Participants) | 0 | 0 | 3 | 0
  CACNA1D c.26_28delAAA |  |  | -33.3 [-79.2 to 41.5] |
  CACNA1D c.58C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CACNA1D c.58C>A |  |  | -33.3 [-79.2 to 41.5] |
  CACNA1I c.2939G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CACNA1I c.2939G>A |  |  | -33.3 [-79.2 to 41.5] |
  CACNA1S c.4718C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CACNA1S c.4718C>T |  |  | 0.0 [-56.1 to 56.1] |
  CAD c.1429G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CAD c.1429G>T |  |  | 33.3 [-41.5 to 79.2] |
  CADPS c.1595G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CADPS c.1595G>A |  |  | -33.3 [-79.2 to 41.5] |
  CAPS2 c.158C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CAPS2 c.158C>T |  |  | -33.3 [-79.2 to 41.5] |
  CARS2 c.1419C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CARS2 c.1419C>T |  |  | -33.3 [-79.2 to 41.5] |
  CATSPERE c.2471A>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  CATSPERE c.2471A>C |  |  | 0.0 [-56.1 to 56.1] |
  CC2D1A c.1030C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CC2D1A c.1030C>T |  |  | -33.3 [-79.2 to 41.5] |
  CC2D2B c.312G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CC2D2B c.312G>A |  |  | -33.3 [-79.2 to 41.5] |
  CCDC105 c.895G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC105 c.895G>A |  |  | -33.3 [-79.2 to 41.5] |
  CCDC114 c.445G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC114 c.445G>A |  |  | -33.3 [-79.2 to 41.5] |
  CCDC142 c.1220G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC142 c.1220G>A |  |  | 0.0 [-56.1 to 56.1] |
  CCDC168 c.17281G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC168 c.17281G>A |  |  | -33.3 [-79.2 to 41.5] |
  CCDC22 c.442C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC22 c.442C>T |  |  | -33.3 [-79.2 to 41.5] |
  CCDC39 c.1189C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC39 c.1189C>G |  |  | 33.3 [-41.5 to 79.2] |
  CCDC47 c.21C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC47 c.21C>A |  |  | 0.0 [-56.1 to 56.1] |
  CCDC70 c.239G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC70 c.239G>A |  |  | -33.3 [-79.2 to 41.5] |
  CCDC73 c.896C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC73 c.896C>T |  |  | -33.3 [-79.2 to 41.5] |
  CCDC8 c.316G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC8 c.316G>A |  |  | 0.0 [-56.1 to 56.1] |
  CCDC91 c.1163C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCDC91 c.1163C>T |  |  | -33.3 [-79.2 to 41.5] |
  CCP110 c.2504G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CCP110 c.2504G>T |  |  | 33.3 [-41.5 to 79.2] |
  CD3G c.497G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CD3G c.497G>A |  |  | -33.3 [-79.2 to 41.5] |
  CD80 c.832G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CD80 c.832G>A |  |  | -33.3 [-79.2 to 41.5] |
  CD9 c.85C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CD9 c.85C>T |  |  | -33.3 [-79.2 to 41.5] |
  CDC25A c.1517G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CDC25A c.1517G>A |  |  | -33.3 [-79.2 to 41.5] |
  CDH13 c.1498G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CDH13 c.1498G>A |  |  | -33.3 [-79.2 to 41.5] |
  CDH23 c.691G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  CDH23 c.691G>C |  |  | 33.3 [-41.5 to 79.2] |
  CDK18 c.1073G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CDK18 c.1073G>A |  |  | -33.3 [-79.2 to 41.5] |
  CDKN2A c.23G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CDKN2A c.23G>A |  |  | -33.3 [-79.2 to 41.5] |
  CDX4 c.455G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CDX4 c.455G>A |  |  | -33.3 [-79.2 to 41.5] |
  CEBPZ c.2155T>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CEBPZ c.2155T>A |  |  | 0.0 [-56.1 to 56.1] |
  CELSR3 c.5802delC: number analyzed (Participants) | 0 | 0 | 3 | 0
  CELSR3 c.5802delC |  |  | 33.3 [-41.5 to 79.2] |
  CELSR3 c.9748C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CELSR3 c.9748C>T |  |  | -33.3 [-79.2 to 41.5] |
  CENPE c.2797G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CENPE c.2797G>A |  |  | -33.3 [-79.2 to 41.5] |
  CENPE c.4270C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CENPE c.4270C>T |  |  | 0.0 [-56.1 to 56.1] |
  CENPV c.596C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CENPV c.596C>T |  |  | -33.3 [-79.2 to 41.5] |
  CEP170B c.1955T>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  CEP170B c.1955T>C |  |  | 33.3 [-41.5 to 79.2] |
  CEP170B c.3520C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  CEP170B c.3520C>G |  |  | -33.3 [-79.2 to 41.5] |
  CEP250 c.589G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CEP250 c.589G>A |  |  | -33.3 [-79.2 to 41.5] |
  CFAP157 c.1441C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CFAP157 c.1441C>A |  |  | -33.3 [-79.2 to 41.5] |
  CFHR4 c.996C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CFHR4 c.996C>A |  |  | -33.3 [-79.2 to 41.5] |
  CGB3 c.427G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CGB3 c.427G>T |  |  | 33.3 [-41.5 to 79.2] |
  CHADL c.868C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CHADL c.868C>A |  |  | 33.3 [-41.5 to 79.2] |
  CHCHD10 c.227G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CHCHD10 c.227G>A |  |  | -33.3 [-79.2 to 41.5] |
  CHD2 c.2366G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CHD2 c.2366G>A |  |  | -33.3 [-79.2 to 41.5] |
  CHD3 c.1796G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CHD3 c.1796G>A |  |  | -33.3 [-79.2 to 41.5] |
  CHD3 c.3880G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CHD3 c.3880G>A |  |  | -33.3 [-79.2 to 41.5] |
  CHPF c.2009A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CHPF c.2009A>T |  |  | 0.0 [-56.1 to 56.1] |
  CHRNA5 c.1192G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CHRNA5 c.1192G>A |  |  | 33.3 [-41.5 to 79.2] |
  CHST13 c.716G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CHST13 c.716G>A |  |  | 33.3 [-41.5 to 79.2] |
  CIZ1 c.626G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CIZ1 c.626G>A |  |  | -33.3 [-79.2 to 41.5] |
  CLCN6 c.698G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CLCN6 c.698G>A |  |  | -33.3 [-79.2 to 41.5] |
  CLCNKA c.476G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CLCNKA c.476G>A |  |  | -33.3 [-79.2 to 41.5] |
  CLDN15 c.301C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CLDN15 c.301C>T |  |  | -33.3 [-79.2 to 41.5] |
  CLEC3A c.547G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CLEC3A c.547G>T |  |  | -33.3 [-79.2 to 41.5] |
  CLEC4F c.839G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CLEC4F c.839G>A |  |  | -33.3 [-79.2 to 41.5] |
  CLIP4 c.890G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  CLIP4 c.890G>C |  |  | -33.3 [-79.2 to 41.5] |
  CLSPN c.533G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CLSPN c.533G>A |  |  | -33.3 [-79.2 to 41.5] |
  CLTA c.698G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CLTA c.698G>A |  |  | 33.3 [-41.5 to 79.2] |
  CLUH c.2743G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CLUH c.2743G>A |  |  | -33.3 [-79.2 to 41.5] |
  CMBL c.460G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CMBL c.460G>A |  |  | 0.0 [-56.1 to 56.1] |
  CNR1 c.982C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CNR1 c.982C>T |  |  | -33.3 [-79.2 to 41.5] |
  CNTD2 c.164C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CNTD2 c.164C>T |  |  | 0.0 [-56.1 to 56.1] |
  COL11A2 c.3100C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  COL11A2 c.3100C>T |  |  | -33.3 [-79.2 to 41.5] |
  COL1A1 c.3680G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  COL1A1 c.3680G>A |  |  | -33.3 [-79.2 to 41.5] |
  COL22A1 c.3584G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  COL22A1 c.3584G>T |  |  | 33.3 [-41.5 to 79.2] |
  COL22A1 c.379C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  COL22A1 c.379C>T |  |  | -33.3 [-79.2 to 41.5] |
  COL27A1 c.2295C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  COL27A1 c.2295C>A |  |  | -33.3 [-79.2 to 41.5] |
  COL4A1 c.3263G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  COL4A1 c.3263G>A |  |  | -33.3 [-79.2 to 41.5] |
  COL6A2 c.1267C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  COL6A2 c.1267C>T |  |  | -33.3 [-79.2 to 41.5] |
  COL6A5 c.5543G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  COL6A5 c.5543G>A |  |  | -33.3 [-79.2 to 41.5] |
  CRB2 c.2873G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CRB2 c.2873G>A |  |  | -33.3 [-79.2 to 41.5] |
  CREB3L1 c.1267C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CREB3L1 c.1267C>T |  |  | -33.3 [-79.2 to 41.5] |
  CRH c.445G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CRH c.445G>A |  |  | -33.3 [-79.2 to 41.5] |
  CRYBG2 c.1418_1419insGTCCCCCACCTGGAAAGAGGTCGTGAAGGGCCCTGGTGCTCCTGCTGCCTC: number analyzed (Participants) | 0 | 0 | 3 | 0
  CRYBG2 c.1418_1419insGTCCCCCACCTGGAAAGAGGTCGTGAAGGGCCCTGGTGCTCCTGCTGCCTC |  |  | 33.3 [-41.5 to 79.2] |
  CSMD1 c.1090G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CSMD1 c.1090G>A |  |  | 0.0 [-56.1 to 56.1] |
  CST9 c.289C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CST9 c.289C>T |  |  | 33.3 [-41.5 to 79.2] |
  CT55 c.331A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CT55 c.331A>T |  |  | 33.3 [-41.5 to 79.2] |
  CTAGE4 c.1963A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  CTAGE4 c.1963A>G |  |  | 33.3 [-41.5 to 79.2] |
  CTBP1 c.1130C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CTBP1 c.1130C>T |  |  | -33.3 [-79.2 to 41.5] |
  CTH c.589C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CTH c.589C>T |  |  | -33.3 [-79.2 to 41.5] |
  CTNNB1 c.1517T>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CTNNB1 c.1517T>A |  |  | 33.3 [-41.5 to 79.2] |
  CTTNBP2 c.3100G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CTTNBP2 c.3100G>A |  |  | 33.3 [-41.5 to 79.2] |
  CX3CL1 c.1130C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  CX3CL1 c.1130C>T |  |  | 33.3 [-41.5 to 79.2] |
  CXCR3 c.386G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CXCR3 c.386G>A |  |  | -33.3 [-79.2 to 41.5] |
  CYBA c.437G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CYBA c.437G>A |  |  | -33.3 [-79.2 to 41.5] |
  CYBB c.1461G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CYBB c.1461G>A |  |  | -33.3 [-79.2 to 41.5] |
  CYGB c.406G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CYGB c.406G>A |  |  | -33.3 [-79.2 to 41.5] |
  CYP2F1 c.1028G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  CYP2F1 c.1028G>A |  |  | 33.3 [-41.5 to 79.2] |
  DAAM1 c.1015C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  DAAM1 c.1015C>T |  |  | -33.3 [-79.2 to 41.5] |
  DAB2 c.2173C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DAB2 c.2173C>A |  |  | 33.3 [-41.5 to 79.2] |
  DACH1 c.1726C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DACH1 c.1726C>A |  |  | -33.3 [-79.2 to 41.5] |
  DALRD3 c.896A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  DALRD3 c.896A>G |  |  | 33.3 [-41.5 to 79.2] |
  DDIAS c.2524G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DDIAS c.2524G>A |  |  | 33.3 [-41.5 to 79.2] |
  DEF8 c.1414G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DEF8 c.1414G>A |  |  | -33.3 [-79.2 to 41.5] |
  DEFB121 c.154G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DEFB121 c.154G>A |  |  | -33.3 [-79.2 to 41.5] |
  DENND1A c.1343G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  DENND1A c.1343G>T |  |  | 0.0 [-56.1 to 56.1] |
  DENND2C c.794G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DENND2C c.794G>A |  |  | -33.3 [-79.2 to 41.5] |
  DENND4A c.311G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DENND4A c.311G>A |  |  | -33.3 [-79.2 to 41.5] |
  DFFB c.379G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DFFB c.379G>A |  |  | -33.3 [-79.2 to 41.5] |
  DGAT1 c.458G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DGAT1 c.458G>A |  |  | -33.3 [-79.2 to 41.5] |
  DGKI c.40C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  DGKI c.40C>T |  |  | -33.3 [-79.2 to 41.5] |
  DHRSX c.721G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DHRSX c.721G>A |  |  | 33.3 [-41.5 to 79.2] |
  DNAH10 c.3640G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DNAH10 c.3640G>A |  |  | -33.3 [-79.2 to 41.5] |
  DNAH9 c.1243C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DNAH9 c.1243C>A |  |  | 33.3 [-41.5 to 79.2] |
  DNAH9 c.6584A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  DNAH9 c.6584A>G |  |  | 33.3 [-41.5 to 79.2] |
  DOCK1 c.5259G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DOCK1 c.5259G>A |  |  | 33.3 [-41.5 to 79.2] |
  DOCK11 c.307G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DOCK11 c.307G>A |  |  | -33.3 [-79.2 to 41.5] |
  DOCK2 c.543C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  DOCK2 c.543C>G |  |  | 0.0 [-56.1 to 56.1] |
  DOCK3 c.2086G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DOCK3 c.2086G>A |  |  | -33.3 [-79.2 to 41.5] |
  DOCK4 c.5740G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  DOCK4 c.5740G>A |  |  | 33.3 [-41.5 to 79.2] |
  DOCK8 c.1205C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  DOCK8 c.1205C>T |  |  | -33.3 [-79.2 to 41.5] |
  DRAM2 c.133G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  DRAM2 c.133G>T |  |  | 33.3 [-41.5 to 79.2] |
  EBPL c.20T>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  EBPL c.20T>C |  |  | -33.3 [-79.2 to 41.5] |
  ECT2 c.619C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ECT2 c.619C>T |  |  | -33.3 [-79.2 to 41.5] |
  EFHC2 c.679G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  EFHC2 c.679G>C |  |  | 0.0 [-56.1 to 56.1] |
  EFHD1 c.88G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  EFHD1 c.88G>T |  |  | 33.3 [-41.5 to 79.2] |
  ELMSAN1 c.939dupC: number analyzed (Participants) | 0 | 0 | 3 | 0
  ELMSAN1 c.939dupC |  |  | 33.3 [-41.5 to 79.2] |
  ELOA2 c.1207G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ELOA2 c.1207G>T |  |  | 33.3 [-41.5 to 79.2] |
  ENC1 c.206G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ENC1 c.206G>A |  |  | 0.0 [-56.1 to 56.1] |
  ENDOG c.142G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ENDOG c.142G>A |  |  | -33.3 [-79.2 to 41.5] |
  ERFE c.467C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ERFE c.467C>T |  |  | -33.3 [-79.2 to 41.5] |
  ESX1 c.959_985delCTGTGCCACCCGGGCCGCCCATGGCGC: number analyzed (Participants) | 0 | 0 | 3 | 0
  ESX1 c.959_985delCTGTGCCACCCGGGCCGCCCATGGCGC |  |  | -33.3 [-79.2 to 41.5] |
  EVC c.1168C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  EVC c.1168C>A |  |  | 33.3 [-41.5 to 79.2] |
  EVC2 c.2095A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  EVC2 c.2095A>G |  |  | 33.3 [-41.5 to 79.2] |
  EVI5 c.1213T>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  EVI5 c.1213T>A |  |  | 33.3 [-41.5 to 79.2] |
  F8 c.3380G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  F8 c.3380G>A |  |  | 33.3 [-41.5 to 79.2] |
  FAAP100 c.22G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAAP100 c.22G>A |  |  | -33.3 [-79.2 to 41.5] |
  FAM135B c.2615G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM135B c.2615G>T |  |  | 33.3 [-41.5 to 79.2] |
  FAM160B2 c.305delC: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM160B2 c.305delC |  |  | 33.3 [-41.5 to 79.2] |
  FAM161B c.932G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM161B c.932G>A |  |  | -33.3 [-79.2 to 41.5] |
  FAM192A c.634C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM192A c.634C>T |  |  | -33.3 [-79.2 to 41.5] |
  FAM210B c.245A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM210B c.245A>G |  |  | 33.3 [-41.5 to 79.2] |
  FAM212A c.216_218delGGA: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM212A c.216_218delGGA |  |  | 33.3 [-41.5 to 79.2] |
  FAM219A c.499G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM219A c.499G>A |  |  | -33.3 [-79.2 to 41.5] |
  FAM220A c.266C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM220A c.266C>T |  |  | 33.3 [-41.5 to 79.2] |
  FAM50B c.307C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM50B c.307C>T |  |  | -33.3 [-79.2 to 41.5] |
  FAM86B2 c.892+5A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM86B2 c.892+5A>G |  |  | 33.3 [-41.5 to 79.2] |
  FAM89A c.110C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FAM89A c.110C>T |  |  | -33.3 [-79.2 to 41.5] |
  FANCA c.4232C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FANCA c.4232C>T |  |  | -33.3 [-79.2 to 41.5] |
  FASN c.4447G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FASN c.4447G>A |  |  | 33.3 [-41.5 to 79.2] |
  FASTKD3 c.20G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FASTKD3 c.20G>A |  |  | -33.3 [-79.2 to 41.5] |
  FBXO3 c.7G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FBXO3 c.7G>A |  |  | -33.3 [-79.2 to 41.5] |
  FBXO33 c.101_109delAGCTGCGAC: number analyzed (Participants) | 0 | 0 | 3 | 0
  FBXO33 c.101_109delAGCTGCGAC |  |  | 33.3 [-41.5 to 79.2] |
  FBXW10 c.1573G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FBXW10 c.1573G>A |  |  | -33.3 [-79.2 to 41.5] |
  FBXW12 c.174A>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  FBXW12 c.174A>C |  |  | 0.0 [-56.1 to 56.1] |
  FBXW9 c.209G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FBXW9 c.209G>A |  |  | 33.3 [-41.5 to 79.2] |
  FCF1 c.589C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FCF1 c.589C>T |  |  | -33.3 [-79.2 to 41.5] |
  FDX1L c.494C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FDX1L c.494C>T |  |  | -33.3 [-79.2 to 41.5] |
  FIGNL2 c.856G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FIGNL2 c.856G>A |  |  | -33.3 [-79.2 to 41.5] |
  FIP1L1 c.1180C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FIP1L1 c.1180C>T |  |  | -33.3 [-79.2 to 41.5] |
  FKBP15 c.3637G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FKBP15 c.3637G>A |  |  | -33.3 [-79.2 to 41.5] |
  FLG c.5378G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FLG c.5378G>A |  |  | 0.0 [-56.1 to 56.1] |
  FLII c.668G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FLII c.668G>A |  |  | -33.3 [-79.2 to 41.5] |
  FLNA c.6100C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FLNA c.6100C>T |  |  | -33.3 [-79.2 to 41.5] |
  FMR1 c.1544G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FMR1 c.1544G>A |  |  | 33.3 [-41.5 to 79.2] |
  FOXD4 c.748_749delGGinsC: number analyzed (Participants) | 0 | 0 | 3 | 0
  FOXD4 c.748_749delGGinsC |  |  | 33.3 [-41.5 to 79.2] |
  FOXN4 c.455delC: number analyzed (Participants) | 0 | 0 | 3 | 0
  FOXN4 c.455delC |  |  | -33.3 [-79.2 to 41.5] |
  FOXO4 c.574C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  FOXO4 c.574C>T |  |  | 0.0 [-56.1 to 56.1] |
  FRAS1 c.5732A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  FRAS1 c.5732A>G |  |  | -33.3 [-79.2 to 41.5] |
  FRS3 c.1336_1344delACCCACCCTinsCCCCCCCCC: number analyzed (Participants) | 0 | 0 | 3 | 0
  FRS3 c.1336_1344delACCCACCCTinsCCCCCCCCC |  |  | 33.3 [-41.5 to 79.2] |
  FSCN2 c.853G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FSCN2 c.853G>A |  |  | -33.3 [-79.2 to 41.5] |
  FSIP2 c.18617_18618delTA: number analyzed (Participants) | 0 | 0 | 3 | 0
  FSIP2 c.18617_18618delTA |  |  | 33.3 [-41.5 to 79.2] |
  FSTL1 c.755G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FSTL1 c.755G>A |  |  | -33.3 [-79.2 to 41.5] |
  FUT7 c.49G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  FUT7 c.49G>A |  |  | -33.3 [-79.2 to 41.5] |
  GAREM1 c.1673G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GAREM1 c.1673G>A |  |  | 0.0 [-56.1 to 56.1] |
  GATAD2B c.1704G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  GATAD2B c.1704G>T |  |  | 33.3 [-41.5 to 79.2] |
  GGCT c.206C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GGCT c.206C>A |  |  | -33.3 [-79.2 to 41.5] |
  GGT5 c.1334C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  GGT5 c.1334C>T |  |  | -33.3 [-79.2 to 41.5] |
  GGT7 c.1093G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GGT7 c.1093G>A |  |  | -33.3 [-79.2 to 41.5] |
  GJA9 c.595G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GJA9 c.595G>A |  |  | -33.3 [-79.2 to 41.5] |
  GLI2 c.4672G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GLI2 c.4672G>A |  |  | 0.0 [-56.1 to 56.1] |
  GLRA4 c.440C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  GLRA4 c.440C>T |  |  | 33.3 [-41.5 to 79.2] |
  GLT8D2 c.278G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GLT8D2 c.278G>A |  |  | -33.3 [-79.2 to 41.5] |
  GMPPB c.887G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GMPPB c.887G>A |  |  | -33.3 [-79.2 to 41.5] |
  GNB1 c.983C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GNB1 c.983C>A |  |  | -33.3 [-79.2 to 41.5] |
  GOLGA2 c.1483C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  GOLGA2 c.1483C>T |  |  | -33.3 [-79.2 to 41.5] |
  GOLGA8K c.1702G>A: number analyzed (Participants) | 0 | 0 | 3 | 2
  GOLGA8K c.1702G>A |  |  | 33.3 [-41.5 to 79.2] | 0.0 [-65.8 to 65.8]
  GOLGA8K c.962A>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  GOLGA8K c.962A>C |  |  | 33.3 [-41.5 to 79.2] |
  GOLIM4 c.949C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  GOLIM4 c.949C>T |  |  | 33.3 [-41.5 to 79.2] |
  GOLM1 c.179G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GOLM1 c.179G>A |  |  | -33.3 [-79.2 to 41.5] |
  GP9 c.131C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  GP9 c.131C>T |  |  | -33.3 [-79.2 to 41.5] |
  GPC1 c.1030G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GPC1 c.1030G>A |  |  | -33.3 [-79.2 to 41.5] |
  GPR149 c.1041C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GPR149 c.1041C>A |  |  | -33.3 [-79.2 to 41.5] |
  GPR155 c.1384G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GPR155 c.1384G>A |  |  | -33.3 [-79.2 to 41.5] |
  GPR50 c.514G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GPR50 c.514G>A |  |  | -33.3 [-79.2 to 41.5] |
  GPR52 c.18G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GPR52 c.18G>A |  |  | -33.3 [-79.2 to 41.5] |
  GPR6 c.715C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  GPR6 c.715C>T |  |  | 33.3 [-41.5 to 79.2] |
  GPR83 c.321C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GPR83 c.321C>A |  |  | -33.3 [-79.2 to 41.5] |
  GPR88 c.568G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GPR88 c.568G>A |  |  | 33.3 [-41.5 to 79.2] |
  GRIA1 c.2318C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  GRIA1 c.2318C>T |  |  | -33.3 [-79.2 to 41.5] |
  GRIA3 c.1913G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GRIA3 c.1913G>A |  |  | -33.3 [-79.2 to 41.5] |
  GRIA3 c.2431G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GRIA3 c.2431G>A |  |  | -33.3 [-79.2 to 41.5] |
  GRK7 c.1027G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GRK7 c.1027G>A |  |  | -33.3 [-79.2 to 41.5] |
  GRK7 c.146G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GRK7 c.146G>A |  |  | 0.0 [-56.1 to 56.1] |
  GRN c.266C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GRN c.266C>A |  |  | -33.3 [-79.2 to 41.5] |
  GSE1 c.1201G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GSE1 c.1201G>A |  |  | -33.3 [-79.2 to 41.5] |
  GSG2 c.611G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GSG2 c.611G>A |  |  | 33.3 [-41.5 to 79.2] |
  GTPBP1 c.1339C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  GTPBP1 c.1339C>T |  |  | 33.3 [-41.5 to 79.2] |
  GUCY2D c.2035G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  GUCY2D c.2035G>A |  |  | -33.3 [-79.2 to 41.5] |
  GYG2 c.910C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  GYG2 c.910C>T |  |  | 0.0 [-56.1 to 56.1] |
  HCFC1 c.4873G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HCFC1 c.4873G>A |  |  | -33.3 [-79.2 to 41.5] |
  HCN1 c.808C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  HCN1 c.808C>T |  |  | -33.3 [-79.2 to 41.5] |
  HDDC2 c.385G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HDDC2 c.385G>A |  |  | -33.3 [-79.2 to 41.5] |
  HDLBP c.1417C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  HDLBP c.1417C>T |  |  | 33.3 [-41.5 to 79.2] |
  HEPHL1 c.3193G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HEPHL1 c.3193G>A |  |  | -33.3 [-79.2 to 41.5] |
  HES2 c.13C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HES2 c.13C>A |  |  | -33.3 [-79.2 to 41.5] |
  HGSNAT c.1622C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  HGSNAT c.1622C>T |  |  | -33.3 [-79.2 to 41.5] |
  HINT3 c.10G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HINT3 c.10G>A |  |  | -33.3 [-79.2 to 41.5] |
  HIP1 c.2956G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HIP1 c.2956G>A |  |  | -33.3 [-79.2 to 41.5] |
  HIST1H2AL c.186G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  HIST1H2AL c.186G>C |  |  | 33.3 [-41.5 to 79.2] |
  HIST2H3D c.19A>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  HIST2H3D c.19A>C |  |  | 33.3 [-41.5 to 79.2] |
  HJURP c.520G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  HJURP c.520G>T |  |  | -33.3 [-79.2 to 41.5] |
  HMGA2 c.275C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  HMGA2 c.275C>T |  |  | 0.0 [-56.1 to 56.1] |
  HNRNPUL2 c.206G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HNRNPUL2 c.206G>A |  |  | -33.3 [-79.2 to 41.5] |
  HOXB9 c.232T>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  HOXB9 c.232T>C |  |  | 33.3 [-41.5 to 79.2] |
  HOXD4 c.121G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HOXD4 c.121G>A |  |  | 33.3 [-41.5 to 79.2] |
  HRG c.988G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HRG c.988G>A |  |  | -33.3 [-79.2 to 41.5] |
  HUNK c.1708C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  HUNK c.1708C>T |  |  | -33.3 [-79.2 to 41.5] |
  HUWE1 c.11869C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HUWE1 c.11869C>A |  |  | 33.3 [-41.5 to 79.2] |
  HYAL3 c.428G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HYAL3 c.428G>A |  |  | -33.3 [-79.2 to 41.5] |
  HYDIN c.10541G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  HYDIN c.10541G>A |  |  | 0.0 [-56.1 to 56.1] |
  ICAM3 c.869G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ICAM3 c.869G>A |  |  | 0.0 [-56.1 to 56.1] |
  IFI30 c.34C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  IFI30 c.34C>T |  |  | 33.3 [-41.5 to 79.2] |
  IFNA10 c.178C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  IFNA10 c.178C>T |  |  | -33.3 [-79.2 to 41.5] |
  IFT81 c.1313G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  IFT81 c.1313G>A |  |  | -33.3 [-79.2 to 41.5] |
  IGFN1 c.5179G>A: number analyzed (Participants) | 0 | 0 | 3 | 2
  IGFN1 c.5179G>A |  |  | 33.3 [-41.5 to 79.2] | -50.0 [-90.5 to 48.6]
  IGFN1 c.5683T>G: number analyzed (Participants) | 0 | 0 | 3 | 2
  IGFN1 c.5683T>G |  |  | 33.3 [-41.5 to 79.2] | 0.0 [-81.1 to 81.1]
  IGFN1 c.5695G>A: number analyzed (Participants) | 0 | 0 | 3 | 2
  IGFN1 c.5695G>A |  |  | 33.3 [-41.5 to 79.2] | 0.0 [-81.1 to 81.1]
  IGSF9B c.932G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  IGSF9B c.932G>A |  |  | -33.3 [-79.2 to 41.5] |
  IL12RB1 c.1097C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  IL12RB1 c.1097C>A |  |  | -33.3 [-79.2 to 41.5] |
  IL6ST c.1165G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  IL6ST c.1165G>A |  |  | -33.3 [-79.2 to 41.5] |
  ILF3 c.1480G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ILF3 c.1480G>A |  |  | 33.3 [-41.5 to 79.2] |
  INA c.41_43delCCT: number analyzed (Participants) | 0 | 0 | 3 | 0
  INA c.41_43delCCT |  |  | -33.3 [-79.2 to 41.5] |
  ING1 c.361C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ING1 c.361C>T |  |  | -33.3 [-79.2 to 41.5] |
  INTS9 c.1412G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  INTS9 c.1412G>A |  |  | -33.3 [-79.2 to 41.5] |
  IQCH c.310C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  IQCH c.310C>T |  |  | -33.3 [-79.2 to 41.5] |
  IQGAP2 c.4025G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  IQGAP2 c.4025G>A |  |  | -33.3 [-79.2 to 41.5] |
  IQSEC3 c.1468G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  IQSEC3 c.1468G>A |  |  | -33.3 [-79.2 to 41.5] |
  ISM2 c.701C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ISM2 c.701C>T |  |  | -33.3 [-79.2 to 41.5] |
  ITGA1 c.3334G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ITGA1 c.3334G>A |  |  | -33.3 [-79.2 to 41.5] |
  ITGA9 c.1040C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ITGA9 c.1040C>T |  |  | -33.3 [-79.2 to 41.5] |
  ITGA9 c.433C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ITGA9 c.433C>T |  |  | -33.3 [-79.2 to 41.5] |
  ITGAE c.1350_1352delGGC: number analyzed (Participants) | 0 | 0 | 3 | 0
  ITGAE c.1350_1352delGGC |  |  | 33.3 [-41.5 to 79.2] |
  ITIH5 c.2035C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ITIH5 c.2035C>T |  |  | -33.3 [-79.2 to 41.5] |
  ITLN2 c.176G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ITLN2 c.176G>A |  |  | -33.3 [-79.2 to 41.5] |
  ITPK1 c.625G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ITPK1 c.625G>A |  |  | -33.3 [-79.2 to 41.5] |
  JMJD7 c.889G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  JMJD7 c.889G>A |  |  | -33.3 [-79.2 to 41.5] |
  JPH3 c.1412C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  JPH3 c.1412C>T |  |  | -33.3 [-79.2 to 41.5] |
  JPH3 c.1688G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  JPH3 c.1688G>A |  |  | -33.3 [-79.2 to 41.5] |
  JSRP1 c.548C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  JSRP1 c.548C>T |  |  | -33.3 [-79.2 to 41.5] |
  KANK3 c.304G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KANK3 c.304G>A |  |  | -33.3 [-79.2 to 41.5] |
  KATNA1 c.443G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KATNA1 c.443G>A |  |  | -33.3 [-79.2 to 41.5] |
  KCNAB3 c.689G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KCNAB3 c.689G>A |  |  | -33.3 [-79.2 to 41.5] |
  KCNE5 c.370C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KCNE5 c.370C>T |  |  | -33.3 [-79.2 to 41.5] |
  KCNG1 c.1226C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KCNG1 c.1226C>T |  |  | -33.3 [-79.2 to 41.5] |
  KCNN4 c.264G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KCNN4 c.264G>T |  |  | 33.3 [-41.5 to 79.2] |
  KCNQ4 c.2041G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KCNQ4 c.2041G>A |  |  | -33.3 [-79.2 to 41.5] |
  KDM2A c.1939G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KDM2A c.1939G>A |  |  | -33.3 [-79.2 to 41.5] |
  KDM6A c.3068G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KDM6A c.3068G>A |  |  | -33.3 [-79.2 to 41.5] |
  KIAA0586 c.397C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIAA0586 c.397C>T |  |  | -33.3 [-79.2 to 41.5] |
  KIAA1109 c.3686C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIAA1109 c.3686C>T |  |  | -33.3 [-79.2 to 41.5] |
  KIAA1324 c.1453G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIAA1324 c.1453G>A |  |  | -33.3 [-79.2 to 41.5] |
  KIF13A c.517C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIF13A c.517C>T |  |  | -33.3 [-79.2 to 41.5] |
  KIF13B c.5231G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIF13B c.5231G>A |  |  | -33.3 [-79.2 to 41.5] |
  KIF17 c.1204G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIF17 c.1204G>A |  |  | 33.3 [-41.5 to 79.2] |
  KIF19 c.92C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIF19 c.92C>T |  |  | -33.3 [-79.2 to 41.5] |
  KIF1B c.2119A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIF1B c.2119A>G |  |  | -33.3 [-79.2 to 41.5] |
  KIF1C c.2522C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIF1C c.2522C>T |  |  | -33.3 [-79.2 to 41.5] |
  KIF21B c.4303G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIF21B c.4303G>A |  |  | 33.3 [-41.5 to 79.2] |
  KIR2DS4 c.436A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KIR2DS4 c.436A>T |  |  | 33.3 [-41.5 to 79.2] |
  KLK2 c.259G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KLK2 c.259G>A |  |  | 33.3 [-41.5 to 79.2] |
  KMT2A c.5755G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KMT2A c.5755G>A |  |  | -33.3 [-79.2 to 41.5] |
  KMT2B c.265G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KMT2B c.265G>A |  |  | -33.3 [-79.2 to 41.5] |
  KNDC1 c.3065C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KNDC1 c.3065C>T |  |  | -33.3 [-79.2 to 41.5] |
  KRBA1 c.1058C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KRBA1 c.1058C>T |  |  | -33.3 [-79.2 to 41.5] |
  KRTAP17-1 c.125G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KRTAP17-1 c.125G>A |  |  | 33.3 [-41.5 to 79.2] |
  KRTAP17-1 c.140G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  KRTAP17-1 c.140G>A |  |  | 33.3 [-41.5 to 79.2] |
  KSR1 c.254C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  KSR1 c.254C>T |  |  | 33.3 [-41.5 to 79.2] |
  LAMA5 c.104C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  LAMA5 c.104C>T |  |  | -33.3 [-79.2 to 41.5] |
  LAMA5 c.7771C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  LAMA5 c.7771C>G |  |  | 0.0 [-56.1 to 56.1] |
  LAMB2 c.2089C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  LAMB2 c.2089C>T |  |  | -33.3 [-79.2 to 41.5] |
  LCE3D c.221G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LCE3D c.221G>A |  |  | 33.3 [-41.5 to 79.2] |
  LDOC1 c.417C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LDOC1 c.417C>A |  |  | -33.3 [-79.2 to 41.5] |
  LEMD3 c.1873C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  LEMD3 c.1873C>T |  |  | -33.3 [-79.2 to 41.5] |
  LINC00452 c.718G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LINC00452 c.718G>A |  |  | 33.3 [-41.5 to 79.2] |
  LIPN c.748A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  LIPN c.748A>G |  |  | -33.3 [-79.2 to 41.5] |
  LKAAEAR1 c.182G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LKAAEAR1 c.182G>A |  |  | -33.3 [-79.2 to 41.5] |
  LMNA c.1634G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LMNA c.1634G>A |  |  | -33.3 [-79.2 to 41.5] |
  LMNA c.356G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LMNA c.356G>A |  |  | -33.3 [-79.2 to 41.5] |
  LMTK3 c.1696G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LMTK3 c.1696G>A |  |  | -33.3 [-79.2 to 41.5] |
  LOC100506388 c.217C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  LOC100506388 c.217C>T |  |  | 33.3 [-41.5 to 79.2] |
  LOC441155 c.35dupT: number analyzed (Participants) | 0 | 0 | 3 | 0
  LOC441155 c.35dupT |  |  | 33.3 [-41.5 to 79.2] |
  LOC729159 c.1004_1005delTGinsCA: number analyzed (Participants) | 0 | 0 | 3 | 0
  LOC729159 c.1004_1005delTGinsCA |  |  | 33.3 [-41.5 to 79.2] |
  LPAR2 c.733A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  LPAR2 c.733A>G |  |  | 33.3 [-41.5 to 79.2] |
  LRP1 c.4006G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LRP1 c.4006G>A |  |  | -33.3 [-79.2 to 41.5] |
  LRRC32 c.1573C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  LRRC32 c.1573C>T |  |  | -33.3 [-79.2 to 41.5] |
  LRRC56 c.899G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LRRC56 c.899G>A |  |  | 33.3 [-41.5 to 79.2] |
  LRRC59 c.510G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  LRRC59 c.510G>C |  |  | 0.0 [-56.1 to 56.1] |
  LRRC8D c.914A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  LRRC8D c.914A>G |  |  | 33.3 [-41.5 to 79.2] |
  LRRN4 c.421A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  LRRN4 c.421A>G |  |  | 33.3 [-41.5 to 79.2] |
  LRRN4 c.442C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  LRRN4 c.442C>T |  |  | 33.3 [-41.5 to 79.2] |
  LYST c.7192G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LYST c.7192G>A |  |  | -33.3 [-79.2 to 41.5] |
  LZTR1 c.1892G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  LZTR1 c.1892G>A |  |  | -33.3 [-79.2 to 41.5] |
  MAD2L2 c.76G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MAD2L2 c.76G>T |  |  | -33.3 [-79.2 to 41.5] |
  MADD c.2251G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MADD c.2251G>A |  |  | 33.3 [-41.5 to 79.2] |
  MAEL c.329T>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  MAEL c.329T>C |  |  | 0.0 [-56.1 to 56.1] |
  MAGEA10 c.145C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MAGEA10 c.145C>T |  |  | -33.3 [-79.2 to 41.5] |
  MAGEA5 c.181C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MAGEA5 c.181C>T |  |  | 0.0 [-56.1 to 56.1] |
  MAGEL2 c.2626G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MAGEL2 c.2626G>A |  |  | 0.0 [-56.1 to 56.1] |
  MAN2A1 c.1916dupA: number analyzed (Participants) | 0 | 0 | 3 | 0
  MAN2A1 c.1916dupA |  |  | -33.3 [-79.2 to 41.5] |
  MANEA c.1096C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MANEA c.1096C>T |  |  | -33.3 [-79.2 to 41.5] |
  MAP7D1 c.2182A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  MAP7D1 c.2182A>G |  |  | 33.3 [-41.5 to 79.2] |
  MARCH1 c.11G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MARCH1 c.11G>T |  |  | -33.3 [-79.2 to 41.5] |
  MARCH2 c.275G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MARCH2 c.275G>T |  |  | 33.3 [-41.5 to 79.2] |
  MAT1A c.280G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  MAT1A c.280G>C |  |  | 33.3 [-41.5 to 79.2] |
  MCCC1 c.667G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MCCC1 c.667G>A |  |  | -33.3 [-79.2 to 41.5] |
  MCM6 c.1693C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MCM6 c.1693C>T |  |  | -33.3 [-79.2 to 41.5] |
  MED12L c.5813C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MED12L c.5813C>T |  |  | -33.3 [-79.2 to 41.5] |
  MED23 c.2836C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MED23 c.2836C>T |  |  | -33.3 [-79.2 to 41.5] |
  MIB2 c.208C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MIB2 c.208C>T |  |  | -33.3 [-79.2 to 41.5] |
  MIER2 c.1453A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  MIER2 c.1453A>G |  |  | 33.3 [-41.5 to 79.2] |
  MIGA2 c.508G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MIGA2 c.508G>A |  |  | -33.3 [-79.2 to 41.5] |
  MIPEP c.1678C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MIPEP c.1678C>T |  |  | -33.3 [-79.2 to 41.5] |
  MLIP c.1145C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MLIP c.1145C>A |  |  | 33.3 [-41.5 to 79.2] |
  MMAB c.733G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MMAB c.733G>A |  |  | -33.3 [-79.2 to 41.5] |
  MMP16 c.391C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MMP16 c.391C>T |  |  | 33.3 [-41.5 to 79.2] |
  MMP24 c.119_121delTGC: number analyzed (Participants) | 0 | 0 | 3 | 0
  MMP24 c.119_121delTGC |  |  | -33.3 [-79.2 to 41.5] |
  MNT c.362C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  MNT c.362C>T |  |  | -33.3 [-79.2 to 41.5] |
  MOV10L1 c.2459A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  MOV10L1 c.2459A>G |  |  | 33.3 [-41.5 to 79.2] |
  MRE11 c.1532delA: number analyzed (Participants) | 0 | 0 | 3 | 0
  MRE11 c.1532delA |  |  | 33.3 [-41.5 to 79.2] |
  MRGPRE c.47G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MRGPRE c.47G>A |  |  | -33.3 [-79.2 to 41.5] |
  MRGPRX4 c.69C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  MRGPRX4 c.69C>G |  |  | 0.0 [-56.1 to 56.1] |
  MROH8 c.598G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MROH8 c.598G>A |  |  | -33.3 [-79.2 to 41.5] |
  MST1R c.931delG: number analyzed (Participants) | 0 | 0 | 3 | 0
  MST1R c.931delG |  |  | -33.3 [-79.2 to 41.5] |
  MTRNR2L3 c.2T>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MTRNR2L3 c.2T>A |  |  | -33.3 [-79.2 to 41.5] |
  MUC12 c.9229C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MUC12 c.9229C>A |  |  | 33.3 [-41.5 to 79.2] |
  MUC16 c.1031G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MUC16 c.1031G>A |  |  | 33.3 [-41.5 to 79.2] |
  MUC19 c.18689G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  MUC19 c.18689G>C |  |  | 33.3 [-41.5 to 79.2] |
  MUC4 c.7666G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MUC4 c.7666G>A |  |  | -33.3 [-79.2 to 41.5] |
  MUC4 c.8866G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MUC4 c.8866G>A |  |  | -33.3 [-79.2 to 41.5] |
  MUT c.1532G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MUT c.1532G>A |  |  | -33.3 [-79.2 to 41.5] |
  MYBPC2 c.3193G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MYBPC2 c.3193G>A |  |  | -33.3 [-79.2 to 41.5] |
  MYH13 c.1440C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  MYH13 c.1440C>G |  |  | 33.3 [-41.5 to 79.2] |
  MYH9 c.4049_4051delAGG: number analyzed (Participants) | 0 | 0 | 3 | 0
  MYH9 c.4049_4051delAGG |  |  | 33.3 [-41.5 to 79.2] |
  MYLK3 c.1105C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  MYLK3 c.1105C>A |  |  | 0.0 [-56.1 to 56.1] |
  MYO7A c.1091delC: number analyzed (Participants) | 0 | 0 | 3 | 0
  MYO7A c.1091delC |  |  | 33.3 [-41.5 to 79.2] |
  NANOS1 c.517G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  NANOS1 c.517G>A |  |  | -33.3 [-79.2 to 41.5] |
  NBPF8 c.1714C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  NBPF8 c.1714C>G |  |  | -33.3 [-79.2 to 41.5] |
  NCAPG2 c.2617C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  NCAPG2 c.2617C>T |  |  | -33.3 [-79.2 to 41.5] |
  NCS1 c.250G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  NCS1 c.250G>A |  |  | -33.3 [-79.2 to 41.5] |
  NEO1 c.3193G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  NEO1 c.3193G>T |  |  | 33.3 [-41.5 to 79.2] |
  NFASC c.1747G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  NFASC c.1747G>A |  |  | 33.3 [-41.5 to 79.2] |
  NISCH c.4270C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  NISCH c.4270C>T |  |  | -33.3 [-79.2 to 41.5] |
  NKX2-5 c.211G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  NKX2-5 c.211G>A |  |  | -33.3 [-79.2 to 41.5] |
  NLGN4X c.166C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  NLGN4X c.166C>T |  |  | -33.3 [-79.2 to 41.5] |
  NLRP3 c.226G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  NLRP3 c.226G>A |  |  | 33.3 [-41.5 to 79.2] |
  NOC2L c.994G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  NOC2L c.994G>A |  |  | -33.3 [-79.2 to 41.5] |
  NOMO2 c.976G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  NOMO2 c.976G>A |  |  | -33.3 [-79.2 to 41.5] |
  NOTCH1 c.1892A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  NOTCH1 c.1892A>G |  |  | -33.3 [-79.2 to 41.5] |
  NPHS1 c.3250delG: number analyzed (Participants) | 0 | 0 | 3 | 0
  NPHS1 c.3250delG |  |  | -33.3 [-79.2 to 41.5] |
  NPTX2 c.979C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  NPTX2 c.979C>T |  |  | -33.3 [-79.2 to 41.5] |
  NTRK2 c.2272G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  NTRK2 c.2272G>A |  |  | -33.3 [-79.2 to 41.5] |
  NUDT16 c.5C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  NUDT16 c.5C>T |  |  | -33.3 [-79.2 to 41.5] |
  NUDT7 c.259G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  NUDT7 c.259G>A |  |  | -33.3 [-79.2 to 41.5] |
  NUDT9 c.480delG: number analyzed (Participants) | 0 | 0 | 3 | 0
  NUDT9 c.480delG |  |  | 33.3 [-41.5 to 79.2] |
  NUFIP1 c.1336G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  NUFIP1 c.1336G>A |  |  | -33.3 [-79.2 to 41.5] |
  NUFIP1 c.415A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  NUFIP1 c.415A>T |  |  | 33.3 [-41.5 to 79.2] |
  NUP210 c.1159C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  NUP210 c.1159C>T |  |  | -33.3 [-79.2 to 41.5] |
  OBSCN c.11180G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  OBSCN c.11180G>A |  |  | -33.3 [-79.2 to 41.5] |
  OBSL1 c.4294C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  OBSL1 c.4294C>T |  |  | -33.3 [-79.2 to 41.5] |
  OGDHL c.2591-11_2600delTGGTCCCTCAGGGACCAGCTT: number analyzed (Participants) | 0 | 0 | 3 | 0
  OGDHL c.2591-11_2600delTGGTCCCTCAGGGACCAGCTT |  |  | -33.3 [-79.2 to 41.5] |
  ONECUT2 c.751C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ONECUT2 c.751C>T |  |  | -33.3 [-79.2 to 41.5] |
  OPRM1 c.266C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  OPRM1 c.266C>T |  |  | 0.0 [-56.1 to 56.1] |
  OR8G5 c.716G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  OR8G5 c.716G>A |  |  | 33.3 [-41.5 to 79.2] |
  OSBPL2 c.543delC: number analyzed (Participants) | 0 | 0 | 3 | 0
  OSBPL2 c.543delC |  |  | 33.3 [-41.5 to 79.2] |
  OVOL1 c.755C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  OVOL1 c.755C>T |  |  | -33.3 [-79.2 to 41.5] |
  PACS2 c.2428G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PACS2 c.2428G>A |  |  | -33.3 [-79.2 to 41.5] |
  PADI2 c.95C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PADI2 c.95C>T |  |  | -33.3 [-79.2 to 41.5] |
  PALD1 c.1525G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PALD1 c.1525G>T |  |  | 33.3 [-41.5 to 79.2] |
  PARD3 c.3457C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PARD3 c.3457C>T |  |  | -33.3 [-79.2 to 41.5] |
  PARS2 c.599G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PARS2 c.599G>A |  |  | -33.3 [-79.2 to 41.5] |
  PCCB c.372G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PCCB c.372G>A |  |  | -33.3 [-79.2 to 41.5] |
  PCDH9 c.3533C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PCDH9 c.3533C>T |  |  | -33.3 [-79.2 to 41.5] |
  PCDH9 c.923C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PCDH9 c.923C>T |  |  | -33.3 [-79.2 to 41.5] |
  PCDHAC2 c.389C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PCDHAC2 c.389C>T |  |  | -33.3 [-79.2 to 41.5] |
  PCDHB13 c.1966G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PCDHB13 c.1966G>A |  |  | -33.3 [-79.2 to 41.5] |
  PCNX3 c.5516_5534delACTGTAGTGGGGGCGGTGG: number analyzed (Participants) | 0 | 0 | 3 | 0
  PCNX3 c.5516_5534delACTGTAGTGGGGGCGGTGG |  |  | 0.0 [-56.1 to 56.1] |
  PCSK4 c.328C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PCSK4 c.328C>T |  |  | -33.3 [-79.2 to 41.5] |
  PCSK5 c.1543A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  PCSK5 c.1543A>G |  |  | 33.3 [-41.5 to 79.2] |
  PDE12 c.806_807delTG: number analyzed (Participants) | 0 | 0 | 3 | 0
  PDE12 c.806_807delTG |  |  | -33.3 [-79.2 to 41.5] |
  PDE1B c.1220C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PDE1B c.1220C>T |  |  | -33.3 [-79.2 to 41.5] |
  PDE1C c.1733G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PDE1C c.1733G>A |  |  | 0.0 [-56.1 to 56.1] |
  PDGFRA c.1365-4C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PDGFRA c.1365-4C>T |  |  | -33.3 [-79.2 to 41.5] |
  PDGFRA c.2645G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PDGFRA c.2645G>A |  |  | -33.3 [-79.2 to 41.5] |
  PDGFRB c.2183+1G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PDGFRB c.2183+1G>A |  |  | -33.3 [-79.2 to 41.5] |
  PDX1 c.172G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  PDX1 c.172G>C |  |  | 33.3 [-41.5 to 79.2] |
  PDZRN3 c.2348C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PDZRN3 c.2348C>T |  |  | 33.3 [-41.5 to 79.2] |
  PELP1 c.2285C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PELP1 c.2285C>T |  |  | -33.3 [-79.2 to 41.5] |
  PGLYRP2 c.1711C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PGLYRP2 c.1711C>T |  |  | -33.3 [-79.2 to 41.5] |
  PHACTR1 c.1248G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PHACTR1 c.1248G>A |  |  | 33.3 [-41.5 to 79.2] |
  PHACTR2 c.1429G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PHACTR2 c.1429G>A |  |  | -33.3 [-79.2 to 41.5] |
  PHF8 c.1499G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PHF8 c.1499G>A |  |  | 33.3 [-41.5 to 79.2] |
  PHF8 c.2385C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PHF8 c.2385C>A |  |  | -33.3 [-79.2 to 41.5] |
  PHLDB1 c.3146G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PHLDB1 c.3146G>A |  |  | -33.3 [-79.2 to 41.5] |
  PHLPP2 c.2843G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PHLPP2 c.2843G>T |  |  | -33.3 [-79.2 to 41.5] |
  PHOX2B c.811C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  PHOX2B c.811C>G |  |  | 33.3 [-41.5 to 79.2] |
  PI4KA c.5701G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PI4KA c.5701G>A |  |  | -33.3 [-79.2 to 41.5] |
  PID1 c.473C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  PID1 c.473C>G |  |  | 33.3 [-41.5 to 79.2] |
  PIDD1 c.992A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  PIDD1 c.992A>G |  |  | 33.3 [-41.5 to 79.2] |
  PIEZO1 c.3107G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PIEZO1 c.3107G>A |  |  | -33.3 [-79.2 to 41.5] |
  PIGG c.1087C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PIGG c.1087C>T |  |  | -33.3 [-79.2 to 41.5] |
  PIGG c.2061G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PIGG c.2061G>A |  |  | -33.3 [-79.2 to 41.5] |
  PIN1 c.220C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PIN1 c.220C>T |  |  | -33.3 [-79.2 to 41.5] |
  PITPNC1 c.527G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PITPNC1 c.527G>T |  |  | 33.3 [-41.5 to 79.2] |
  PKHD1 c.5814G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PKHD1 c.5814G>T |  |  | -33.3 [-79.2 to 41.5] |
  PLCB1 c.2279G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PLCB1 c.2279G>A |  |  | 33.3 [-41.5 to 79.2] |
  PLEK2 c.458G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PLEK2 c.458G>A |  |  | -33.3 [-79.2 to 41.5] |
  PLEKHA5 c.1070C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PLEKHA5 c.1070C>T |  |  | -33.3 [-79.2 to 41.5] |
  PLEKHG1 c.2273G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PLEKHG1 c.2273G>A |  |  | -33.3 [-79.2 to 41.5] |
  PLEKHM1 c.2174G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PLEKHM1 c.2174G>A |  |  | -33.3 [-79.2 to 41.5] |
  PLK5 c.505C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PLK5 c.505C>T |  |  | 0.0 [-56.1 to 56.1] |
  PLXNB1 c.4699G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PLXNB1 c.4699G>A |  |  | -33.3 [-79.2 to 41.5] |
  PNPT1 c.1285-3_1288delAAGTTTCinsTTTTTTT: number analyzed (Participants) | 0 | 0 | 3 | 0
  PNPT1 c.1285-3_1288delAAGTTTCinsTTTTTTT |  |  | 33.3 [-41.5 to 79.2] |
  PODXL2 c.1217G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PODXL2 c.1217G>A |  |  | -33.3 [-79.2 to 41.5] |
  POLR2A c.1492G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  POLR2A c.1492G>A |  |  | -33.3 [-79.2 to 41.5] |
  POM121C c.1456A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  POM121C c.1456A>T |  |  | 33.3 [-41.5 to 79.2] |
  POMT1 c.1648C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  POMT1 c.1648C>T |  |  | 33.3 [-41.5 to 79.2] |
  POTEF c.505C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  POTEF c.505C>A |  |  | 33.3 [-41.5 to 79.2] |
  POU3F3 c.259G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  POU3F3 c.259G>A |  |  | 0.0 [-56.1 to 56.1] |
  PPEF1 c.735C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PPEF1 c.735C>A |  |  | -33.3 [-79.2 to 41.5] |
  PRAMEF11 c.1144A>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  PRAMEF11 c.1144A>C |  |  | -33.3 [-79.2 to 41.5] |
  PREP c.815G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PREP c.815G>A |  |  | -33.3 [-79.2 to 41.5] |
  PRR14L c.3470A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  PRR14L c.3470A>G |  |  | 33.3 [-41.5 to 79.2] |
  PRSS55 c.43G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PRSS55 c.43G>A |  |  | 33.3 [-41.5 to 79.2] |
  PTPRS c.2192C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  PTPRS c.2192C>T |  |  | -33.3 [-79.2 to 41.5] |
  PTPRS c.2872C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  PTPRS c.2872C>A |  |  | -33.3 [-79.2 to 41.5] |
  QRICH2 c.3259G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  QRICH2 c.3259G>A |  |  | -33.3 [-79.2 to 41.5] |
  QSOX2 c.994C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  QSOX2 c.994C>T |  |  | -33.3 [-79.2 to 41.5] |
  R3HCC1 c.309-1G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  R3HCC1 c.309-1G>A |  |  | 33.3 [-41.5 to 79.2] |
  RAB21 c.41_43delCGG: number analyzed (Participants) | 0 | 0 | 3 | 0
  RAB21 c.41_43delCGG |  |  | -33.3 [-79.2 to 41.5] |
  RAD50 c.1684G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RAD50 c.1684G>A |  |  | -33.3 [-79.2 to 41.5] |
  RAD54L2 c.1012A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  RAD54L2 c.1012A>G |  |  | -33.3 [-79.2 to 41.5] |
  RALGAPA2 c.1332G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RALGAPA2 c.1332G>T |  |  | -33.3 [-79.2 to 41.5] |
  RAPH1 c.1993G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RAPH1 c.1993G>A |  |  | -33.3 [-79.2 to 41.5] |
  RASAL3 c.2062G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RASAL3 c.2062G>A |  |  | 33.3 [-41.5 to 79.2] |
  RASAL3 c.2155G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  RASAL3 c.2155G>C |  |  | 33.3 [-41.5 to 79.2] |
  RASGRF2 c.123G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  RASGRF2 c.123G>C |  |  | 33.3 [-41.5 to 79.2] |
  RASGRP4 c.1501G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RASGRP4 c.1501G>A |  |  | -33.3 [-79.2 to 41.5] |
  RB1 c.2359C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RB1 c.2359C>T |  |  | -33.3 [-79.2 to 41.5] |
  RBL1 c.294A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RBL1 c.294A>T |  |  | 33.3 [-41.5 to 79.2] |
  RBM25 c.1438G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RBM25 c.1438G>A |  |  | -33.3 [-79.2 to 41.5] |
  RBM43 c.167C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RBM43 c.167C>T |  |  | -33.3 [-79.2 to 41.5] |
  RBMXL3 c.1307G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RBMXL3 c.1307G>A |  |  | -33.3 [-79.2 to 41.5] |
  RBPMS c.50A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  RBPMS c.50A>G |  |  | 0.0 [-56.1 to 56.1] |
  RFPL2 c.1018_1021delTTGCinsCTGT: number analyzed (Participants) | 0 | 0 | 3 | 0
  RFPL2 c.1018_1021delTTGCinsCTGT |  |  | 33.3 [-41.5 to 79.2] |
  RFPL2 c.970A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  RFPL2 c.970A>G |  |  | 33.3 [-41.5 to 79.2] |
  RGPD3 c.2468A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RGPD3 c.2468A>T |  |  | 33.3 [-41.5 to 79.2] |
  RGS20 c.1145C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RGS20 c.1145C>T |  |  | -33.3 [-79.2 to 41.5] |
  RIMS4 c.597G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RIMS4 c.597G>T |  |  | 33.3 [-41.5 to 79.2] |
  RIMS4 c.730G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  RIMS4 c.730G>C |  |  | 0.0 [-56.1 to 56.1] |
  RIOK3 c.1010C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RIOK3 c.1010C>T |  |  | -33.3 [-79.2 to 41.5] |
  RNASEL c.1419A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RNASEL c.1419A>T |  |  | 0.0 [-56.1 to 56.1] |
  RNF114 c.680A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RNF114 c.680A>T |  |  | 33.3 [-41.5 to 79.2] |
  RNF123 c.3932C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RNF123 c.3932C>T |  |  | 33.3 [-41.5 to 79.2] |
  RNF185 c.254G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RNF185 c.254G>A |  |  | -33.3 [-79.2 to 41.5] |
  RNF185 c.558G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RNF185 c.558G>A |  |  | -33.3 [-79.2 to 41.5] |
  RNF214 c.412G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RNF214 c.412G>A |  |  | -33.3 [-79.2 to 41.5] |
  RNH1 c.433G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RNH1 c.433G>T |  |  | -33.3 [-79.2 to 41.5] |
  RPAP3 c.1011delA: number analyzed (Participants) | 0 | 0 | 3 | 0
  RPAP3 c.1011delA |  |  | -33.3 [-79.2 to 41.5] |
  RPL18 c.335G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RPL18 c.335G>A |  |  | 33.3 [-41.5 to 79.2] |
  RPL4 c.427C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RPL4 c.427C>T |  |  | -33.3 [-79.2 to 41.5] |
  RPS6KA2 c.1756G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RPS6KA2 c.1756G>A |  |  | -33.3 [-79.2 to 41.5] |
  RPS6KB2 c.37G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RPS6KB2 c.37G>A |  |  | 33.3 [-41.5 to 79.2] |
  RRBP1 c.2335G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RRBP1 c.2335G>A |  |  | -33.3 [-79.2 to 41.5] |
  RTN1 c.1600C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RTN1 c.1600C>A |  |  | 0.0 [-56.1 to 56.1] |
  RTP5 c.281G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  RTP5 c.281G>A |  |  | -33.3 [-79.2 to 41.5] |
  RUNDC1 c.337C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RUNDC1 c.337C>T |  |  | 33.3 [-41.5 to 79.2] |
  RXFP2 c.604C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  RXFP2 c.604C>T |  |  | -33.3 [-79.2 to 41.5] |
  SACS c.2488G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SACS c.2488G>A |  |  | -33.3 [-79.2 to 41.5] |
  SALL3 c.1837G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SALL3 c.1837G>A |  |  | -33.3 [-79.2 to 41.5] |
  SAMHD1 c.405_421delCATTGATACACCTCAAT: number analyzed (Participants) | 0 | 0 | 3 | 0
  SAMHD1 c.405_421delCATTGATACACCTCAAT |  |  | 0.0 [-56.1 to 56.1] |
  SAP30L c.193G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SAP30L c.193G>A |  |  | -33.3 [-79.2 to 41.5] |
  SAPCD1 c.119G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SAPCD1 c.119G>A |  |  | -33.3 [-79.2 to 41.5] |
  SBSN c.1583A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SBSN c.1583A>T |  |  | 0.0 [-56.1 to 56.1] |
  SCAP c.2892delC: number analyzed (Participants) | 0 | 0 | 3 | 0
  SCAP c.2892delC |  |  | 33.3 [-41.5 to 79.2] |
  SEC14L1 c.1129C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SEC14L1 c.1129C>T |  |  | -33.3 [-79.2 to 41.5] |
  SEC14L4 c.287G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SEC14L4 c.287G>T |  |  | -33.3 [-79.2 to 41.5] |
  SEC24D c.907G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SEC24D c.907G>A |  |  | -33.3 [-79.2 to 41.5] |
  SH2D3C c.898C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SH2D3C c.898C>T |  |  | 33.3 [-41.5 to 79.2] |
  SIGLEC9 c.17_19delTGC: number analyzed (Participants) | 0 | 0 | 3 | 0
  SIGLEC9 c.17_19delTGC |  |  | 33.3 [-41.5 to 79.2] |
  SIRPG c.1141G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SIRPG c.1141G>A |  |  | -33.3 [-79.2 to 41.5] |
  SLC22A8 c.583G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC22A8 c.583G>A |  |  | -33.3 [-79.2 to 41.5] |
  SLC26A4 c.575T>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC26A4 c.575T>C |  |  | -33.3 [-79.2 to 41.5] |
  SLC2A5 c.964G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC2A5 c.964G>A |  |  | -33.3 [-79.2 to 41.5] |
  SLC2A6 c.961G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC2A6 c.961G>A |  |  | -33.3 [-79.2 to 41.5] |
  SLC2A8 c.576delC: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC2A8 c.576delC |  |  | -33.3 [-79.2 to 41.5] |
  SLC35F1 c.703G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC35F1 c.703G>A |  |  | 0.0 [-56.1 to 56.1] |
  SLC44A3 c.332A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC44A3 c.332A>T |  |  | -33.3 [-79.2 to 41.5] |
  SLC5A10 c.1211G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC5A10 c.1211G>A |  |  | -33.3 [-79.2 to 41.5] |
  SLC6A13 c.1341C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC6A13 c.1341C>A |  |  | -33.3 [-79.2 to 41.5] |
  SLC8A1 c.2011A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC8A1 c.2011A>T |  |  | 0.0 [-56.1 to 56.1] |
  SLC8A3 c.2374G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLC8A3 c.2374G>A |  |  | -33.3 [-79.2 to 41.5] |
  SLIT3 c.182G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SLIT3 c.182G>A |  |  | -33.3 [-79.2 to 41.5] |
  SMARCA4 c.4185delA: number analyzed (Participants) | 0 | 0 | 3 | 0
  SMARCA4 c.4185delA |  |  | 33.3 [-41.5 to 79.2] |
  SMARCAD1 c.1637G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SMARCAD1 c.1637G>A |  |  | -33.3 [-79.2 to 41.5] |
  SOBP c.1950G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SOBP c.1950G>T |  |  | -33.3 [-79.2 to 41.5] |
  SOGA1 c.1477G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SOGA1 c.1477G>T |  |  | 0.0 [-56.1 to 56.1] |
  SOST c.278C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SOST c.278C>A |  |  | 33.3 [-41.5 to 79.2] |
  SOX18 c.698C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SOX18 c.698C>T |  |  | -33.3 [-79.2 to 41.5] |
  SP140 c.2167G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SP140 c.2167G>A |  |  | -33.3 [-79.2 to 41.5] |
  SP8 c.326G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SP8 c.326G>A |  |  | -33.3 [-79.2 to 41.5] |
  SPATA31A6 c.1997A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  SPATA31A6 c.1997A>G |  |  | 33.3 [-41.5 to 79.2] |
  SPATA31E1 c.2987G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SPATA31E1 c.2987G>A |  |  | -33.3 [-79.2 to 41.5] |
  SPINK2 c.118A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  SPINK2 c.118A>G |  |  | 33.3 [-41.5 to 79.2] |
  SPIRE2 c.470_472delAGG: number analyzed (Participants) | 0 | 0 | 3 | 0
  SPIRE2 c.470_472delAGG |  |  | -33.3 [-79.2 to 41.5] |
  SPOCD1 c.3199G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SPOCD1 c.3199G>A |  |  | -33.3 [-79.2 to 41.5] |
  SREBF2 c.85G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SREBF2 c.85G>A |  |  | -33.3 [-79.2 to 41.5] |
  SSC4D c.1154C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SSC4D c.1154C>T |  |  | 33.3 [-41.5 to 79.2] |
  SSH2 c.2626G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  SSH2 c.2626G>C |  |  | 0.0 [-56.1 to 56.1] |
  SSPO c.13487A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  SSPO c.13487A>G |  |  | 33.3 [-41.5 to 79.2] |
  SSPO c.1967G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SSPO c.1967G>T |  |  | -33.3 [-79.2 to 41.5] |
  SSTR1 c.121C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SSTR1 c.121C>T |  |  | -33.3 [-79.2 to 41.5] |
  STAC3 c.226_227insGGG: number analyzed (Participants) | 0 | 0 | 3 | 0
  STAC3 c.226_227insGGG |  |  | -33.3 [-79.2 to 41.5] |
  STK26 c.1073C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  STK26 c.1073C>T |  |  | -33.3 [-79.2 to 41.5] |
  STK33 c.1280G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  STK33 c.1280G>C |  |  | 33.3 [-41.5 to 79.2] |
  STK38L c.148G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  STK38L c.148G>A |  |  | -33.3 [-79.2 to 41.5] |
  STK40 c.1198G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  STK40 c.1198G>A |  |  | 33.3 [-41.5 to 79.2] |
  STT3B c.957T>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  STT3B c.957T>G |  |  | 33.3 [-41.5 to 79.2] |
  SUDS3 c.397_399delAAG: number analyzed (Participants) | 0 | 0 | 3 | 0
  SUDS3 c.397_399delAAG |  |  | 33.3 [-41.5 to 79.2] |
  SUSD3 c.428C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SUSD3 c.428C>T |  |  | -33.3 [-79.2 to 41.5] |
  SYCP2 c.4180C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  SYCP2 c.4180C>T |  |  | -33.3 [-79.2 to 41.5] |
  SYN2 c.544G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SYN2 c.544G>A |  |  | -33.3 [-79.2 to 41.5] |
  SYNE2 c.9263G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  SYNE2 c.9263G>A |  |  | 33.3 [-41.5 to 79.2] |
  TACC2 c.2488C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  TACC2 c.2488C>T |  |  | 33.3 [-41.5 to 79.2] |
  TACC2 c.3196G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TACC2 c.3196G>A |  |  | 33.3 [-41.5 to 79.2] |
  TACC3 c.1847C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  TACC3 c.1847C>T |  |  | -33.3 [-79.2 to 41.5] |
  TAF1D c.281delA: number analyzed (Participants) | 0 | 0 | 3 | 0
  TAF1D c.281delA |  |  | 33.3 [-41.5 to 79.2] |
  TBL1X c.826C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  TBL1X c.826C>T |  |  | 33.3 [-41.5 to 79.2] |
  TEKT4 c.824G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TEKT4 c.824G>A |  |  | -33.3 [-79.2 to 41.5] |
  TET1 c.5408G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TET1 c.5408G>A |  |  | -33.3 [-79.2 to 41.5] |
  TEX264 c.875G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TEX264 c.875G>A |  |  | 33.3 [-41.5 to 79.2] |
  TFAP2E c.305C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  TFAP2E c.305C>T |  |  | -33.3 [-79.2 to 41.5] |
  TFRC c.1763G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TFRC c.1763G>A |  |  | -33.3 [-79.2 to 41.5] |
  TGM4 c.937G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TGM4 c.937G>A |  |  | 33.3 [-41.5 to 79.2] |
  THEMIS2 c.1527_1531delTGTGAinsCGTGG: number analyzed (Participants) | 0 | 0 | 3 | 0
  THEMIS2 c.1527_1531delTGTGAinsCGTGG |  |  | 33.3 [-41.5 to 79.2] |
  TIGD4 c.373G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TIGD4 c.373G>A |  |  | -33.3 [-79.2 to 41.5] |
  TLN1 c.7088C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  TLN1 c.7088C>T |  |  | 33.3 [-41.5 to 79.2] |
  TMC6 c.2054G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMC6 c.2054G>A |  |  | -33.3 [-79.2 to 41.5] |
  TMCO6 c.464T>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMCO6 c.464T>A |  |  | 0.0 [-56.1 to 56.1] |
  TMEM151A c.3G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMEM151A c.3G>A |  |  | 33.3 [-41.5 to 79.2] |
  TMEM165 c.703C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMEM165 c.703C>G |  |  | 33.3 [-41.5 to 79.2] |
  TMEM200B c.338G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMEM200B c.338G>T |  |  | 33.3 [-41.5 to 79.2] |
  TMEM232 c.1045G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMEM232 c.1045G>A |  |  | -33.3 [-79.2 to 41.5] |
  TMEM237 c.1159G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMEM237 c.1159G>A |  |  | -33.3 [-79.2 to 41.5] |
  TMEM59L c.800G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMEM59L c.800G>A |  |  | 33.3 [-41.5 to 79.2] |
  TMEM63C c.2128C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMEM63C c.2128C>T |  |  | -33.3 [-79.2 to 41.5] |
  TMEM70 c.113G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMEM70 c.113G>T |  |  | -33.3 [-79.2 to 41.5] |
  TMEM94 c.859G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TMEM94 c.859G>A |  |  | -33.3 [-79.2 to 41.5] |
  TNFSF18 c.355A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  TNFSF18 c.355A>G |  |  | -33.3 [-79.2 to 41.5] |
  TNRC18 c.3076A>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  TNRC18 c.3076A>C |  |  | 33.3 [-41.5 to 79.2] |
  TNRC6B c.4934G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TNRC6B c.4934G>A |  |  | 0.0 [-56.1 to 56.1] |
  TOGARAM1 c.2390A>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  TOGARAM1 c.2390A>C |  |  | 0.0 [-56.1 to 56.1] |
  TOP2B c.1057C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  TOP2B c.1057C>G |  |  | 0.0 [-56.1 to 56.1] |
  TOP2B c.247G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TOP2B c.247G>A |  |  | -33.3 [-79.2 to 41.5] |
  TPR c.583A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  TPR c.583A>G |  |  | 0.0 [-56.1 to 56.1] |
  TRDN c.1900G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TRDN c.1900G>A |  |  | -33.3 [-79.2 to 41.5] |
  TRIM61 c.365C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  TRIM61 c.365C>G |  |  | 33.3 [-41.5 to 79.2] |
  TRIM64B c.377delG: number analyzed (Participants) | 0 | 0 | 3 | 0
  TRIM64B c.377delG |  |  | 33.3 [-41.5 to 79.2] |
  TRPV1 c.1753A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  TRPV1 c.1753A>G |  |  | 33.3 [-41.5 to 79.2] |
  TSEN2 c.247C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  TSEN2 c.247C>G |  |  | 0.0 [-56.1 to 56.1] |
  TSEN2 c.451G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TSEN2 c.451G>A |  |  | 0.0 [-56.1 to 56.1] |
  TSEN2 c.506G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TSEN2 c.506G>A |  |  | 0.0 [-56.1 to 56.1] |
  TTK c.1324_1327delTCTA: number analyzed (Participants) | 0 | 0 | 3 | 0
  TTK c.1324_1327delTCTA |  |  | 33.3 [-41.5 to 79.2] |
  TTN c.68658G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  TTN c.68658G>C |  |  | 33.3 [-41.5 to 79.2] |
  TTN c.68716C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TTN c.68716C>A |  |  | -33.3 [-79.2 to 41.5] |
  TTPA c.103G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  TTPA c.103G>A |  |  | 33.3 [-41.5 to 79.2] |
  TULP4 c.4571C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  TULP4 c.4571C>T |  |  | -33.3 [-79.2 to 41.5] |
  TXNRD2 c.1522C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  TXNRD2 c.1522C>T |  |  | -33.3 [-79.2 to 41.5] |
  UBASH3B c.32G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  UBASH3B c.32G>A |  |  | -33.3 [-79.2 to 41.5] |
  UBE4A c.2306G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  UBE4A c.2306G>A |  |  | -33.3 [-79.2 to 41.5] |
  USP32 c.2804G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  USP32 c.2804G>A |  |  | -33.3 [-79.2 to 41.5] |
  USPL1 c.3256G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  USPL1 c.3256G>A |  |  | -33.3 [-79.2 to 41.5] |
  VGLL2 c.794C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  VGLL2 c.794C>T |  |  | -33.3 [-79.2 to 41.5] |
  WDFY3 c.1262T>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  WDFY3 c.1262T>C |  |  | 0.0 [-56.1 to 56.1] |
  WDR18 c.1075C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  WDR18 c.1075C>A |  |  | 33.3 [-41.5 to 79.2] |
  XKR4 c.1918A>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  XKR4 c.1918A>T |  |  | 33.3 [-41.5 to 79.2] |
  XPO4 c.238C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  XPO4 c.238C>T |  |  | -33.3 [-79.2 to 41.5] |
  XPO7 c.2398C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  XPO7 c.2398C>T |  |  | -33.3 [-79.2 to 41.5] |
  ZAR1 c.1145C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZAR1 c.1145C>T |  |  | -33.3 [-79.2 to 41.5] |
  ZC3H12B c.2285G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZC3H12B c.2285G>A |  |  | -33.3 [-79.2 to 41.5] |
  ZC3H12D c.1213C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZC3H12D c.1213C>T |  |  | 33.3 [-41.5 to 79.2] |
  ZC3H7B c.1569C>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZC3H7B c.1569C>G |  |  | 33.3 [-41.5 to 79.2] |
  ZC3H8 c.220G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZC3H8 c.220G>A |  |  | -33.3 [-79.2 to 41.5] |
  ZDBF2 c.5228C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZDBF2 c.5228C>T |  |  | 33.3 [-41.5 to 79.2] |
  ZMPSTE24 c.1085dupT: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZMPSTE24 c.1085dupT |  |  | -33.3 [-79.2 to 41.5] |
  ZMYM1 c.1965G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZMYM1 c.1965G>A |  |  | -33.3 [-79.2 to 41.5] |
  ZMYM5 c.74C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZMYM5 c.74C>T |  |  | -33.3 [-79.2 to 41.5] |
  ZMYND15 c.1468G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZMYND15 c.1468G>A |  |  | -33.3 [-79.2 to 41.5] |
  ZNF10 c.1658C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF10 c.1658C>T |  |  | 0.0 [-56.1 to 56.1] |
  ZNF207 c.673A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF207 c.673A>G |  |  | 33.3 [-41.5 to 79.2] |
  ZNF208 c.766T>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF208 c.766T>C |  |  | -33.3 [-79.2 to 41.5] |
  ZNF276 c.548C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF276 c.548C>T |  |  | -33.3 [-79.2 to 41.5] |
  ZNF365 c.307G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF365 c.307G>A |  |  | 0.0 [-56.1 to 56.1] |
  ZNF367 c.854G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF367 c.854G>A |  |  | 33.3 [-41.5 to 79.2] |
  ZNF37A c.1369C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF37A c.1369C>T |  |  | 33.3 [-41.5 to 79.2] |
  ZNF383 c.820C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF383 c.820C>T |  |  | -33.3 [-79.2 to 41.5] |
  ZNF420 c.34G>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF420 c.34G>T |  |  | -33.3 [-79.2 to 41.5] |
  ZNF431 c.1260G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF431 c.1260G>A |  |  | -33.3 [-79.2 to 41.5] |
  ZNF431 c.1462G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF431 c.1462G>A |  |  | -33.3 [-79.2 to 41.5] |
  ZNF431 c.1525G>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF431 c.1525G>C |  |  | -33.3 [-79.2 to 41.5] |
  ZNF474 c.757C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF474 c.757C>T |  |  | 0.0 [-56.1 to 56.1] |
  ZNF493 c.802G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF493 c.802G>A |  |  | -33.3 [-79.2 to 41.5] |
  ZNF536 c.3551A>C: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF536 c.3551A>C |  |  | 33.3 [-41.5 to 79.2] |
  ZNF568 c.1066C>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF568 c.1066C>A |  |  | 0.0 [-56.1 to 56.1] |
  ZNF680 c.1016A>G: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF680 c.1016A>G |  |  | -33.3 [-79.2 to 41.5] |
  ZNF696 c.430C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF696 c.430C>T |  |  | 33.3 [-41.5 to 79.2] |
  ZNF782 c.1630G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNF782 c.1630G>A |  |  | -33.3 [-79.2 to 41.5] |
  ZNFX1 c.1982C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZNFX1 c.1982C>T |  |  | -33.3 [-79.2 to 41.5] |
  ZP1 c.1103G>A: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZP1 c.1103G>A |  |  | -33.3 [-79.2 to 41.5] |
  ZYX c.697C>T: number analyzed (Participants) | 0 | 0 | 3 | 0
  ZYX c.697C>T |  |  | -33.3 [-79.2 to 41.5] |
  ABCA5 c.725_727delCAGinsAAA: number analyzed (Participants) | 0 | 0 | 0 | 2
  ABCA5 c.725_727delCAGinsAAA |  |  |  | 50.0 [-48.6 to 90.5]
  ACSF3 c.1180C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ACSF3 c.1180C>A |  |  |  | -50.0 [-90.5 to 48.6]
  ADAMTS2 c.2243C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  ADAMTS2 c.2243C>T |  |  |  | -50.0 [-90.5 to 48.6]
  ADCK2 c.253C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  ADCK2 c.253C>T |  |  |  | 0.0 [-65.8 to 65.8]
  ADGRA1 c.227G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ADGRA1 c.227G>A |  |  |  | -50.0 [-90.5 to 48.6]
  ADGRF3 c.1615G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ADGRF3 c.1615G>A |  |  |  | -50.0 [-90.5 to 48.6]
  ADGRG2 c.1314C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ADGRG2 c.1314C>A |  |  |  | -50.0 [-90.5 to 48.6]
  ADGRV1 c.16006C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ADGRV1 c.16006C>A |  |  |  | -50.0 [-90.5 to 48.6]
  AFAP1 c.140A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  AFAP1 c.140A>G |  |  |  | -50.0 [-90.5 to 48.6]
  AHNAK c.14273A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  AHNAK c.14273A>G |  |  |  | 0.0 [-65.8 to 65.8]
  AHRR c.1881C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  AHRR c.1881C>A |  |  |  | 0.0 [-65.8 to 65.8]
  AKAP13 c.5222C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  AKAP13 c.5222C>A |  |  |  | -50.0 [-90.5 to 48.6]
  AKR1B15 c.452delT: number analyzed (Participants) | 0 | 0 | 0 | 2
  AKR1B15 c.452delT |  |  |  | -50.0 [-90.5 to 48.6]
  ALS2CR12 c.1079C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ALS2CR12 c.1079C>A |  |  |  | -50.0 [-90.5 to 48.6]
  ALX3 c.226G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ALX3 c.226G>A |  |  |  | -50.0 [-90.5 to 48.6]
  AMOTL2 c.2426G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  AMOTL2 c.2426G>A |  |  |  | -50.0 [-90.5 to 48.6]
  ANK3 c.9349dupA: number analyzed (Participants) | 0 | 0 | 0 | 2
  ANK3 c.9349dupA |  |  |  | -50.0 [-90.5 to 48.6]
  ANKRD33 c.112G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ANKRD33 c.112G>A |  |  |  | -50.0 [-90.5 to 48.6]
  ANXA10 c.655G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  ANXA10 c.655G>T |  |  |  | -50.0 [-90.5 to 48.6]
  AP4B1 c.1657G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  AP4B1 c.1657G>A |  |  |  | 50.0 [-48.6 to 90.5]
  APPBP2 c.863C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  APPBP2 c.863C>A |  |  |  | 50.0 [-48.6 to 90.5]
  ARHGAP6 c.1393G>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  ARHGAP6 c.1393G>C |  |  |  | 0.0 [-65.8 to 65.8]
  ARID1A c.492_494delCGC: number analyzed (Participants) | 0 | 0 | 0 | 2
  ARID1A c.492_494delCGC |  |  |  | -50.0 [-90.5 to 48.6]
  ARMC12 c.829G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ARMC12 c.829G>A |  |  |  | 0.0 [-65.8 to 65.8]
  ARSE c.1750C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ARSE c.1750C>A |  |  |  | -50.0 [-90.5 to 48.6]
  ATM c.458G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  ATM c.458G>T |  |  |  | -50.0 [-90.5 to 48.6]
  ATM c.6889C>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  ATM c.6889C>G |  |  |  | -50.0 [-90.5 to 48.6]
  ATP10D c.545G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  ATP10D c.545G>T |  |  |  | -50.0 [-90.5 to 48.6]
  ATXN3 c.911_912insACAGCAGCAGCAGCAGCAGCAGCA: number analyzed (Participants) | 0 | 0 | 0 | 2
  ATXN3 c.911_912insACAGCAGCAGCAGCAGCAGCAGCA |  |  |  | -50.0 [-90.5 to 48.6]
  ATXN7 c.59_61delCGG: number analyzed (Participants) | 0 | 0 | 0 | 2
  ATXN7 c.59_61delCGG |  |  |  | 50.0 [-48.6 to 90.5]
  BCR c.3055G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  BCR c.3055G>A |  |  |  | -50.0 [-90.5 to 48.6]
  BRIX1 c.494T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  BRIX1 c.494T>C |  |  |  | -50.0 [-90.5 to 48.6]
  BTG2 c.17G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  BTG2 c.17G>A |  |  |  | 50.0 [-48.6 to 90.5]
  C10orf76 c.1715T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  C10orf76 c.1715T>C |  |  |  | 0.0 [-65.8 to 65.8]
  C10orf82 c.343G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  C10orf82 c.343G>T |  |  |  | -50.0 [-90.5 to 48.6]
  C10orf95 c.581G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  C10orf95 c.581G>A |  |  |  | -50.0 [-90.5 to 48.6]
  C12orf56 c.989A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  C12orf56 c.989A>G |  |  |  | -50.0 [-90.5 to 48.6]
  C16orf86 c.922C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  C16orf86 c.922C>T |  |  |  | -50.0 [-90.5 to 48.6]
  C3 c.641C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  C3 c.641C>A |  |  |  | -50.0 [-90.5 to 48.6]
  CACFD1 c.665_668delCCCT: number analyzed (Participants) | 0 | 0 | 0 | 2
  CACFD1 c.665_668delCCCT |  |  |  | -50.0 [-90.5 to 48.6]
  CAMKK2 c.1599_1601delGACinsAACAAAA: number analyzed (Participants) | 0 | 0 | 0 | 2
  CAMKK2 c.1599_1601delGACinsAACAAAA |  |  |  | 50.0 [-48.6 to 90.5]
  CAPN13 c.1888A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  CAPN13 c.1888A>G |  |  |  | -50.0 [-90.5 to 48.6]
  CASKIN2 c.3538A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  CASKIN2 c.3538A>G |  |  |  | -50.0 [-90.5 to 48.6]
  CASQ2 c.51C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CASQ2 c.51C>A |  |  |  | -50.0 [-90.5 to 48.6]
  CCDC106 c.138G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CCDC106 c.138G>T |  |  |  | -50.0 [-90.5 to 48.6]
  CCDC114 c.601A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  CCDC114 c.601A>G |  |  |  | 50.0 [-48.6 to 90.5]
  CCDC144A c.1001C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CCDC144A c.1001C>A |  |  |  | -50.0 [-90.5 to 48.6]
  CCDC168 c.15025G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CCDC168 c.15025G>A |  |  |  | -50.0 [-90.5 to 48.6]
  CCDC25 c.137C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CCDC25 c.137C>A |  |  |  | -50.0 [-90.5 to 48.6]
  CCDC93 c.1321G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CCDC93 c.1321G>T |  |  |  | -50.0 [-90.5 to 48.6]
  CCNI2 c.460G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CCNI2 c.460G>A |  |  |  | 0.0 [-65.8 to 65.8]
  CCNL2 c.532A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  CCNL2 c.532A>G |  |  |  | 0.0 [-65.8 to 65.8]
  CCT3 c.591delA: number analyzed (Participants) | 0 | 0 | 0 | 2
  CCT3 c.591delA |  |  |  | -50.0 [-90.5 to 48.6]
  CD1B c.418G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CD1B c.418G>T |  |  |  | -50.0 [-90.5 to 48.6]
  CD7 c.44C>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  CD7 c.44C>G |  |  |  | -50.0 [-90.5 to 48.6]
  CDH17 c.1315G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CDH17 c.1315G>A |  |  |  | -50.0 [-90.5 to 48.6]
  CDK6 c.631G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CDK6 c.631G>A |  |  |  | -50.0 [-90.5 to 48.6]
  CECR2 c.3651_3655dupAACCC: number analyzed (Participants) | 0 | 0 | 0 | 2
  CECR2 c.3651_3655dupAACCC |  |  |  | 0.0 [-65.8 to 65.8]
  CELSR1 c.5418G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CELSR1 c.5418G>T |  |  |  | -50.0 [-90.5 to 48.6]
  CEP128 c.3073G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CEP128 c.3073G>T |  |  |  | -50.0 [-90.5 to 48.6]
  CEP290 c.5517G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CEP290 c.5517G>T |  |  |  | -50.0 [-90.5 to 48.6]
  CEP85L c.11G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CEP85L c.11G>T |  |  |  | -50.0 [-90.5 to 48.6]
  CFAP36 c.685G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CFAP36 c.685G>A |  |  |  | -50.0 [-90.5 to 48.6]
  CFAP53 c.984_988delGAAACinsAAAAA: number analyzed (Participants) | 0 | 0 | 0 | 2
  CFAP53 c.984_988delGAAACinsAAAAA |  |  |  | 50.0 [-48.6 to 90.5]
  CFAP65 c.2247G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CFAP65 c.2247G>A |  |  |  | -50.0 [-90.5 to 48.6]
  CFAP97 c.481delA: number analyzed (Participants) | 0 | 0 | 0 | 2
  CFAP97 c.481delA |  |  |  | -50.0 [-90.5 to 48.6]
  CGB3 c.16-2A>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CGB3 c.16-2A>T |  |  |  | 50.0 [-48.6 to 90.5]
  CHEK2 c.1409A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  CHEK2 c.1409A>G |  |  |  | -50.0 [-90.5 to 48.6]
  CIZ1 c.346C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CIZ1 c.346C>A |  |  |  | -50.0 [-90.5 to 48.6]
  CLCN1 c.2435_2445delAGCCTGTCTGT: number analyzed (Participants) | 0 | 0 | 0 | 2
  CLCN1 c.2435_2445delAGCCTGTCTGT |  |  |  | 50.0 [-48.6 to 90.5]
  CLCN3 c.1469G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CLCN3 c.1469G>A |  |  |  | -50.0 [-90.5 to 48.6]
  CLDN19 c.503G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CLDN19 c.503G>A |  |  |  | -50.0 [-90.5 to 48.6]
  CLEC18C c.299T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  CLEC18C c.299T>C |  |  |  | -50.0 [-90.5 to 48.6]
  CLN5 c.272C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CLN5 c.272C>T |  |  |  | -50.0 [-90.5 to 48.6]
  CLPTM1L c.1295T>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CLPTM1L c.1295T>A |  |  |  | 0.0 [-65.8 to 65.8]
  CNOT1 c.4630_4635delCTGTTAinsTTTTTT: number analyzed (Participants) | 0 | 0 | 0 | 2
  CNOT1 c.4630_4635delCTGTTAinsTTTTTT |  |  |  | -50.0 [-90.5 to 48.6]
  CNTN6 c.2759G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CNTN6 c.2759G>A |  |  |  | -50.0 [-90.5 to 48.6]
  COL11A2 c.2102C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  COL11A2 c.2102C>T |  |  |  | -50.0 [-90.5 to 48.6]
  COL19A1 c.1703G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  COL19A1 c.1703G>A |  |  |  | -50.0 [-90.5 to 48.6]
  COL27A1 c.1908G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  COL27A1 c.1908G>A |  |  |  | 50.0 [-48.6 to 90.5]
  CP c.2291C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CP c.2291C>T |  |  |  | -50.0 [-90.5 to 48.6]
  CPB2 c.340delC: number analyzed (Participants) | 0 | 0 | 0 | 2
  CPB2 c.340delC |  |  |  | 50.0 [-48.6 to 90.5]
  CRYBG3 c.4646C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CRYBG3 c.4646C>A |  |  |  | 0.0 [-65.8 to 65.8]
  CXCL6 c.86C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  CXCL6 c.86C>T |  |  |  | -50.0 [-90.5 to 48.6]
  CXorf36 c.587G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CXorf36 c.587G>A |  |  |  | -50.0 [-90.5 to 48.6]
  CYP11B2 c.1471C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  CYP11B2 c.1471C>A |  |  |  | -50.0 [-90.5 to 48.6]
  DCC c.601C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  DCC c.601C>T |  |  |  | 50.0 [-48.6 to 90.5]
  DEPDC1B c.682G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  DEPDC1B c.682G>A |  |  |  | 0.0 [-65.8 to 65.8]
  DHRS2 c.287A>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  DHRS2 c.287A>T |  |  |  | 0.0 [-65.8 to 65.8]
  DHX29 c.3296C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  DHX29 c.3296C>A |  |  |  | -50.0 [-90.5 to 48.6]
  DLG5 c.2296G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  DLG5 c.2296G>T |  |  |  | -50.0 [-90.5 to 48.6]
  DNAAF3 c.976G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  DNAAF3 c.976G>A |  |  |  | 0.0 [-65.8 to 65.8]
  DNAH9 c.6762G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  DNAH9 c.6762G>T |  |  |  | -50.0 [-90.5 to 48.6]
  DOLPP1 c.500A>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  DOLPP1 c.500A>T |  |  |  | -50.0 [-90.5 to 48.6]
  DSC2 c.934G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  DSC2 c.934G>T |  |  |  | 0.0 [-65.8 to 65.8]
  DST c.4384G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  DST c.4384G>T |  |  |  | 0.0 [-65.8 to 65.8]
  EML5 c.824G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  EML5 c.824G>A |  |  |  | 0.0 [-65.8 to 65.8]
  ENAM c.869G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ENAM c.869G>A |  |  |  | -50.0 [-90.5 to 48.6]
  ENO4 c.1751A>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  ENO4 c.1751A>T |  |  |  | 50.0 [-48.6 to 90.5]
  ENPEP c.1552G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  ENPEP c.1552G>T |  |  |  | -50.0 [-90.5 to 48.6]
  EOGT c.419C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  EOGT c.419C>T |  |  |  | -50.0 [-90.5 to 48.6]
  EPG5 c.6263T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  EPG5 c.6263T>G |  |  |  | -50.0 [-90.5 to 48.6]
  EREG c.143G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  EREG c.143G>A |  |  |  | 0.0 [-65.8 to 65.8]
  ESRP2 c.381G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ESRP2 c.381G>A |  |  |  | -50.0 [-90.5 to 48.6]
  EXOSC10 c.1751C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  EXOSC10 c.1751C>T |  |  |  | 50.0 [-48.6 to 90.5]
  F13A1 c.1909-883_2038dup: number analyzed (Participants) | 0 | 0 | 0 | 2
  F13A1 c.1909-883_2038dup |  |  |  | -50.0 [-90.5 to 48.6]
  F2RL1 c.280G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  F2RL1 c.280G>A |  |  |  | -50.0 [-90.5 to 48.6]
  FAM186A c.4757_4828delAACTGGGGATCCCTCTCACCCCTCAGC AGGCGCAGGAACTGGGGATCCCTCTCACCCCTCAGCAGGC GCAGG: number analyzed (Participants) | 0 | 0 | 0 | 2
  FAM186A c.4757_4828delAACTGGGGATCCCTCTCACCCCTCAGC AGGCGCAGGAACTGGGGATCCCTCTCACCCCTCAGCAGGC GCAGG |  |  |  | 50.0 [-48.6 to 90.5]
  FAM193A c.1769C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  FAM193A c.1769C>T |  |  |  | -50.0 [-90.5 to 48.6]
  FAM90A1 c.1261G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  FAM90A1 c.1261G>T |  |  |  | 50.0 [-48.6 to 90.5]
  FAM9B c.285G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  FAM9B c.285G>T |  |  |  | -50.0 [-90.5 to 48.6]
  FANCI c.153C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  FANCI c.153C>A |  |  |  | -50.0 [-90.5 to 48.6]
  FARSB c.1177C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  FARSB c.1177C>T |  |  |  | 50.0 [-48.6 to 90.5]
  FAT1 c.10630G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  FAT1 c.10630G>A |  |  |  | -50.0 [-90.5 to 48.6]
  FBL c.407C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  FBL c.407C>T |  |  |  | -50.0 [-90.5 to 48.6]
  FGF10 c.365C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  FGF10 c.365C>T |  |  |  | -50.0 [-90.5 to 48.6]
  FIG4 c.2347G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  FIG4 c.2347G>A |  |  |  | 50.0 [-48.6 to 90.5]
  FIG4 c.2586A>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  FIG4 c.2586A>T |  |  |  | 0.0 [-65.8 to 65.8]
  FNTA c.408C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  FNTA c.408C>A |  |  |  | -50.0 [-90.5 to 48.6]
  FOXRED1 c.104C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  FOXRED1 c.104C>T |  |  |  | -50.0 [-90.5 to 48.6]
  FOXRED1 c.65G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  FOXRED1 c.65G>A |  |  |  | -50.0 [-90.5 to 48.6]
  FXR2 c.994A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  FXR2 c.994A>G |  |  |  | -50.0 [-90.5 to 48.6]
  GAB3 c.1307C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GAB3 c.1307C>A |  |  |  | -50.0 [-90.5 to 48.6]
  GAGE2A c.175C>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  GAGE2A c.175C>G |  |  |  | 50.0 [-48.6 to 90.5]
  GALR2 c.646C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GALR2 c.646C>A |  |  |  | -50.0 [-90.5 to 48.6]
  GDF7 c.955C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  GDF7 c.955C>T |  |  |  | -50.0 [-90.5 to 48.6]
  GFRA1 c.665C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  GFRA1 c.665C>T |  |  |  | -50.0 [-90.5 to 48.6]
  GGT1 c.1081G>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  GGT1 c.1081G>C |  |  |  | -50.0 [-90.5 to 48.6]
  GHR c.1705C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GHR c.1705C>A |  |  |  | -50.0 [-90.5 to 48.6]
  GIPR c.301C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  GIPR c.301C>T |  |  |  | -50.0 [-90.5 to 48.6]
  GKAP1 c.424G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GKAP1 c.424G>A |  |  |  | 50.0 [-48.6 to 90.5]
  GKAP1 c.427G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GKAP1 c.427G>A |  |  |  | 50.0 [-48.6 to 90.5]
  GKAP1 c.432C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GKAP1 c.432C>A |  |  |  | 50.0 [-48.6 to 90.5]
  GLP1R c.16G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  GLP1R c.16G>T |  |  |  | -50.0 [-90.5 to 48.6]
  GLYATL2 c.680A>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  GLYATL2 c.680A>C |  |  |  | -50.0 [-90.5 to 48.6]
  GLYATL2 c.705A>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  GLYATL2 c.705A>C |  |  |  | -50.0 [-90.5 to 48.6]
  GLYR1 c.1120G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GLYR1 c.1120G>A |  |  |  | -50.0 [-90.5 to 48.6]
  GMNN c.161G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GMNN c.161G>A |  |  |  | -50.0 [-90.5 to 48.6]
  GNRH2 c.40_42delCTG: number analyzed (Participants) | 0 | 0 | 0 | 2
  GNRH2 c.40_42delCTG |  |  |  | -50.0 [-90.5 to 48.6]
  GOLGA8A c.1463C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  GOLGA8A c.1463C>T |  |  |  | 50.0 [-48.6 to 90.5]
  GOLGA8A c.1505G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GOLGA8A c.1505G>A |  |  |  | 50.0 [-48.6 to 90.5]
  GOLGA8A c.1538G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GOLGA8A c.1538G>A |  |  |  | 0.0 [-65.8 to 65.8]
  GRIK4 c.2590C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  GRIK4 c.2590C>T |  |  |  | 0.0 [-65.8 to 65.8]
  GRM7 c.2014G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  GRM7 c.2014G>A |  |  |  | -50.0 [-90.5 to 48.6]
  H2AFY c.10C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  H2AFY c.10C>T |  |  |  | 0.0 [-65.8 to 65.8]
  HAUS5 c.425C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  HAUS5 c.425C>T |  |  |  | -50.0 [-90.5 to 48.6]
  HERC1 c.11036G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  HERC1 c.11036G>A |  |  |  | 50.0 [-48.6 to 90.5]
  HIF3A c.1573C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  HIF3A c.1573C>T |  |  |  | 0.0 [-65.8 to 65.8]
  HOXA13 c.396_398delCGC: number analyzed (Participants) | 0 | 0 | 0 | 2
  HOXA13 c.396_398delCGC |  |  |  | 50.0 [-48.6 to 90.5]
  HOXD13 c.120C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  HOXD13 c.120C>A |  |  |  | -50.0 [-90.5 to 48.6]
  HRH1 c.1048C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  HRH1 c.1048C>A |  |  |  | 50.0 [-48.6 to 90.5]
  HRNR c.7688G>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  HRNR c.7688G>C |  |  |  | 50.0 [-48.6 to 90.5]
  HSD17B12 c.682C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  HSD17B12 c.682C>T |  |  |  | -50.0 [-90.5 to 48.6]
  HSPG2 c.8873C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  HSPG2 c.8873C>T |  |  |  | -50.0 [-90.5 to 48.6]
  HUWE1 c.1553C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  HUWE1 c.1553C>A |  |  |  | -50.0 [-90.5 to 48.6]
  HUWE1 c.1924G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  HUWE1 c.1924G>T |  |  |  | -50.0 [-90.5 to 48.6]
  HUWE1 c.7633C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  HUWE1 c.7633C>A |  |  |  | -50.0 [-90.5 to 48.6]
  ICAM4 c.38dupT: number analyzed (Participants) | 0 | 0 | 0 | 2
  ICAM4 c.38dupT |  |  |  | -50.0 [-90.5 to 48.6]
  IGFN1 c.5612A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  IGFN1 c.5612A>G |  |  |  | -50.0 [-90.5 to 48.6]
  IGFN1 c.5624C>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  IGFN1 c.5624C>G |  |  |  | 0.0 [-65.8 to 65.8]
  IL12RB1 c.1442G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  IL12RB1 c.1442G>A |  |  |  | -50.0 [-90.5 to 48.6]
  ILF2 c.40_41delGGinsTT: number analyzed (Participants) | 0 | 0 | 0 | 2
  ILF2 c.40_41delGGinsTT |  |  |  | 0.0 [-65.8 to 65.8]
  IQSEC3 c.973G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  IQSEC3 c.973G>A |  |  |  | 0.0 [-65.8 to 65.8]
  ITGAD c.2240G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ITGAD c.2240G>A |  |  |  | 0.0 [-65.8 to 65.8]
  ITPR2 c.8022G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  ITPR2 c.8022G>T |  |  |  | -50.0 [-90.5 to 48.6]
  JKAMP c.158G>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  JKAMP c.158G>C |  |  |  | 0.0 [-65.8 to 65.8]
  JPH3 c.169A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  JPH3 c.169A>G |  |  |  | -50.0 [-90.5 to 48.6]
  KIAA0513 c.646G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  KIAA0513 c.646G>T |  |  |  | -50.0 [-90.5 to 48.6]
  KIAA0895 c.720C>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  KIAA0895 c.720C>G |  |  |  | 0.0 [-65.8 to 65.8]
  KIAA1107 c.3152C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  KIAA1107 c.3152C>A |  |  |  | -50.0 [-90.5 to 48.6]
  KIAA1107 c.3310C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  KIAA1107 c.3310C>A |  |  |  | -50.0 [-90.5 to 48.6]
  KIF5C c.226G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  KIF5C c.226G>T |  |  |  | -50.0 [-90.5 to 48.6]
  KLHL34 c.1513G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  KLHL34 c.1513G>T |  |  |  | -50.0 [-90.5 to 48.6]
  KLHL9 c.825T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  KLHL9 c.825T>G |  |  |  | 0.0 [-65.8 to 65.8]
  KLRK1 c.197G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  KLRK1 c.197G>A |  |  |  | 50.0 [-48.6 to 90.5]
  KMT5C c.1141dupC: number analyzed (Participants) | 0 | 0 | 0 | 2
  KMT5C c.1141dupC |  |  |  | -50.0 [-90.5 to 48.6]
  KNL1 c.1800G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  KNL1 c.1800G>T |  |  |  | -50.0 [-90.5 to 48.6]
  KRT13 c.610G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  KRT13 c.610G>A |  |  |  | 0.0 [-65.8 to 65.8]
  KRTAP9-9 c.35_36insACCTGCTGCAGGACC: number analyzed (Participants) | 0 | 0 | 0 | 2
  KRTAP9-9 c.35_36insACCTGCTGCAGGACC |  |  |  | 50.0 [-48.6 to 90.5]
  LCA5L c.1198G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  LCA5L c.1198G>A |  |  |  | 50.0 [-48.6 to 90.5]
  LCAT c.625C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  LCAT c.625C>A |  |  |  | -50.0 [-90.5 to 48.6]
  LCT c.1925C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  LCT c.1925C>A |  |  |  | -50.0 [-90.5 to 48.6]
  LDB3 c.2012G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  LDB3 c.2012G>A |  |  |  | -50.0 [-90.5 to 48.6]
  LILRB5 c.1274C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  LILRB5 c.1274C>T |  |  |  | -50.0 [-90.5 to 48.6]
  LMNA c.1977G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  LMNA c.1977G>T |  |  |  | -50.0 [-90.5 to 48.6]
  LMO7 c.1315T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  LMO7 c.1315T>C |  |  |  | 50.0 [-48.6 to 90.5]
  LOC100505841 c.50G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  LOC100505841 c.50G>A |  |  |  | -50.0 [-90.5 to 48.6]
  LOC101928841 c.3272G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  LOC101928841 c.3272G>A |  |  |  | -50.0 [-90.5 to 48.6]
  LONRF3 c.712C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  LONRF3 c.712C>A |  |  |  | -50.0 [-90.5 to 48.6]
  LRP2 c.13139dupC: number analyzed (Participants) | 0 | 0 | 0 | 2
  LRP2 c.13139dupC |  |  |  | -50.0 [-90.5 to 48.6]
  LRRC4 c.912_913delTG: number analyzed (Participants) | 0 | 0 | 0 | 2
  LRRC4 c.912_913delTG |  |  |  | 50.0 [-48.6 to 90.5]
  LRRC40 c.1457C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  LRRC40 c.1457C>T |  |  |  | 50.0 [-48.6 to 90.5]
  LRRK1 c.644G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  LRRK1 c.644G>A |  |  |  | -50.0 [-90.5 to 48.6]
  LTBP1 c.307C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  LTBP1 c.307C>T |  |  |  | -50.0 [-90.5 to 48.6]
  MADD c.3458C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  MADD c.3458C>T |  |  |  | -50.0 [-90.5 to 48.6]
  MAP2K2 c.1069C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  MAP2K2 c.1069C>T |  |  |  | -50.0 [-90.5 to 48.6]
  MAZ c.272C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  MAZ c.272C>T |  |  |  | 50.0 [-48.6 to 90.5]
  MED21 c.35T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  MED21 c.35T>G |  |  |  | 0.0 [-65.8 to 65.8]
  MED23 c.2276dupA: number analyzed (Participants) | 0 | 0 | 0 | 2
  MED23 c.2276dupA |  |  |  | -50.0 [-90.5 to 48.6]
  METTL5 c.388G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  METTL5 c.388G>A |  |  |  | 0.0 [-65.8 to 65.8]
  MICALL1 c.2475C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MICALL1 c.2475C>A |  |  |  | -50.0 [-90.5 to 48.6]
  MIER3 c.1113delG: number analyzed (Participants) | 0 | 0 | 0 | 2
  MIER3 c.1113delG |  |  |  | 0.0 [-65.8 to 65.8]
  MMP2 c.1484G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MMP2 c.1484G>A |  |  |  | -50.0 [-90.5 to 48.6]
  MMP24 c.170_172delCGG: number analyzed (Participants) | 0 | 0 | 0 | 2
  MMP24 c.170_172delCGG |  |  |  | 50.0 [-48.6 to 90.5]
  MRPL21 c.581G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MRPL21 c.581G>A |  |  |  | 0.0 [-65.8 to 65.8]
  MRVI1 c.1446delA: number analyzed (Participants) | 0 | 0 | 0 | 2
  MRVI1 c.1446delA |  |  |  | -50.0 [-90.5 to 48.6]
  MUC12 c.13432C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC12 c.13432C>A |  |  |  | 50.0 [-48.6 to 90.5]
  MUC12 c.2740T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC12 c.2740T>C |  |  |  | 50.0 [-48.6 to 90.5]
  MUC12 c.4291G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC12 c.4291G>A |  |  |  | 50.0 [-48.6 to 90.5]
  MUC12 c.5251A>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC12 c.5251A>C |  |  |  | 0.0 [-65.8 to 65.8]
  MUC12 c.5512C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC12 c.5512C>A |  |  |  | 50.0 [-48.6 to 90.5]
  MUC12 c.5575G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC12 c.5575G>A |  |  |  | 50.0 [-48.6 to 90.5]
  MUC12 c.5612C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC12 c.5612C>T |  |  |  | 50.0 [-48.6 to 90.5]
  MUC16 c.17447G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC16 c.17447G>A |  |  |  | 0.0 [-65.8 to 65.8]
  MUC19 c.3641G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC19 c.3641G>A |  |  |  | 0.0 [-65.8 to 65.8]
  MUC4 c.3605T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC4 c.3605T>C |  |  |  | 50.0 [-48.6 to 90.5]
  MUC4 c.7039A>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC4 c.7039A>T |  |  |  | 50.0 [-48.6 to 90.5]
  MUC4 c.8259_10034dup: number analyzed (Participants) | 0 | 0 | 0 | 2
  MUC4 c.8259_10034dup |  |  |  | 50.0 [-48.6 to 90.5]
  MVD c.665G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MVD c.665G>A |  |  |  | -50.0 [-90.5 to 48.6]
  MX1 c.454G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MX1 c.454G>A |  |  |  | 50.0 [-48.6 to 90.5]
  MYCBP2 c.1826C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  MYCBP2 c.1826C>T |  |  |  | -50.0 [-90.5 to 48.6]
  MYCBP2 c.3572C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  MYCBP2 c.3572C>T |  |  |  | -50.0 [-90.5 to 48.6]
  MYH14 c.2935G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  MYH14 c.2935G>A |  |  |  | 0.0 [-65.8 to 65.8]
  MYOF c.1772_1773delAG: number analyzed (Participants) | 0 | 0 | 0 | 2
  MYOF c.1772_1773delAG |  |  |  | -50.0 [-90.5 to 48.6]
  MYOM3 c.221C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  MYOM3 c.221C>T |  |  |  | -50.0 [-90.5 to 48.6]
  NALCN c.2063_2065delCCT: number analyzed (Participants) | 0 | 0 | 0 | 2
  NALCN c.2063_2065delCCT |  |  |  | 0.0 [-65.8 to 65.8]
  NANOGNB c.495_501delGCATAAGinsAAAAAAA: number analyzed (Participants) | 0 | 0 | 0 | 2
  NANOGNB c.495_501delGCATAAGinsAAAAAAA |  |  |  | 50.0 [-48.6 to 90.5]
  NBEA c.5218G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  NBEA c.5218G>T |  |  |  | 50.0 [-48.6 to 90.5]
  NCKIPSD c.1430C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  NCKIPSD c.1430C>T |  |  |  | 50.0 [-48.6 to 90.5]
  NEB c.17635-2_17635delAGAinsTTT: number analyzed (Participants) | 0 | 0 | 0 | 2
  NEB c.17635-2_17635delAGAinsTTT |  |  |  | -50.0 [-90.5 to 48.6]
  NEK1 c.739C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  NEK1 c.739C>T |  |  |  | -50.0 [-90.5 to 48.6]
  NEPRO c.837delA: number analyzed (Participants) | 0 | 0 | 0 | 2
  NEPRO c.837delA |  |  |  | -50.0 [-90.5 to 48.6]
  NEUROD6 c.89A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  NEUROD6 c.89A>G |  |  |  | -50.0 [-90.5 to 48.6]
  NFATC1 c.179C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  NFATC1 c.179C>T |  |  |  | -50.0 [-90.5 to 48.6]
  NHS c.2203C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  NHS c.2203C>T |  |  |  | -50.0 [-90.5 to 48.6]
  NLRP12 c.2971C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  NLRP12 c.2971C>A |  |  |  | -50.0 [-90.5 to 48.6]
  NLRP14 c.3228G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  NLRP14 c.3228G>T |  |  |  | -50.0 [-90.5 to 48.6]
  NLRP6 c.176C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  NLRP6 c.176C>T |  |  |  | -50.0 [-90.5 to 48.6]
  NMD3 c.754G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  NMD3 c.754G>T |  |  |  | -50.0 [-90.5 to 48.6]
  NPHP3 c.1525-4_1526delCTAGTAinsTTTTTT: number analyzed (Participants) | 0 | 0 | 0 | 2
  NPHP3 c.1525-4_1526delCTAGTAinsTTTTTT |  |  |  | 50.0 [-48.6 to 90.5]
  NR2E1 c.592C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  NR2E1 c.592C>A |  |  |  | -50.0 [-90.5 to 48.6]
  NRAP c.4058G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  NRAP c.4058G>T |  |  |  | -50.0 [-90.5 to 48.6]
  NRG2 c.2084G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  NRG2 c.2084G>A |  |  |  | -50.0 [-90.5 to 48.6]
  NUCB1 c.664C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  NUCB1 c.664C>T |  |  |  | -50.0 [-90.5 to 48.6]
  NUP98 c.2972C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  NUP98 c.2972C>A |  |  |  | -50.0 [-90.5 to 48.6]
  NYAP2 c.703G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  NYAP2 c.703G>A |  |  |  | 0.0 [-65.8 to 65.8]
  NYNRIN c.3662G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  NYNRIN c.3662G>A |  |  |  | 0.0 [-65.8 to 65.8]
  OBSCN c.6543G>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  OBSCN c.6543G>C |  |  |  | 0.0 [-65.8 to 65.8]
  OR13C5 c.243_244delGC: number analyzed (Participants) | 0 | 0 | 0 | 2
  OR13C5 c.243_244delGC |  |  |  | 50.0 [-48.6 to 90.5]
  OR2T2 c.612_618delCGTGCTG: number analyzed (Participants) | 0 | 0 | 0 | 2
  OR2T2 c.612_618delCGTGCTG |  |  |  | 0.0 [-65.8 to 65.8]
  OR2T2 c.785T>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  OR2T2 c.785T>A |  |  |  | 50.0 [-48.6 to 90.5]
  OR2T3 c.611T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  OR2T3 c.611T>C |  |  |  | 50.0 [-48.6 to 90.5]
  OR2T8 c.590T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  OR2T8 c.590T>G |  |  |  | -50.0 [-90.5 to 48.6]
  OR2W3 c.337C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  OR2W3 c.337C>A |  |  |  | -50.0 [-90.5 to 48.6]
  OR4C12 c.222_224delTTC: number analyzed (Participants) | 0 | 0 | 0 | 2
  OR4C12 c.222_224delTTC |  |  |  | -50.0 [-90.5 to 48.6]
  OR51A4 c.497_500delGAAAinsCAAG: number analyzed (Participants) | 0 | 0 | 0 | 2
  OR51A4 c.497_500delGAAAinsCAAG |  |  |  | 50.0 [-48.6 to 90.5]
  OR52D1 c.127G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  OR52D1 c.127G>T |  |  |  | 50.0 [-48.6 to 90.5]
  OSMR c.937G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  OSMR c.937G>T |  |  |  | -50.0 [-90.5 to 48.6]
  OTOF c.5567G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  OTOF c.5567G>A |  |  |  | -50.0 [-90.5 to 48.6]
  PADI3 c.1739C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  PADI3 c.1739C>A |  |  |  | -50.0 [-90.5 to 48.6]
  PCDH18 c.809C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  PCDH18 c.809C>T |  |  |  | -50.0 [-90.5 to 48.6]
  PCDH8 c.1583G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  PCDH8 c.1583G>A |  |  |  | -50.0 [-90.5 to 48.6]
  PCLO c.2545G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  PCLO c.2545G>A |  |  |  | 0.0 [-65.8 to 65.8]
  PGLYRP3 c.551G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  PGLYRP3 c.551G>T |  |  |  | 0.0 [-65.8 to 65.8]
  PGS1 c.1069A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  PGS1 c.1069A>G |  |  |  | 0.0 [-65.8 to 65.8]
  PIGO c.3116delT: number analyzed (Participants) | 0 | 0 | 0 | 2
  PIGO c.3116delT |  |  |  | 0.0 [-65.8 to 65.8]
  PKD1 c.2647C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  PKD1 c.2647C>A |  |  |  | -50.0 [-90.5 to 48.6]
  PLD3 c.464C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  PLD3 c.464C>T |  |  |  | 0.0 [-65.8 to 65.8]
  PLK2 c.328G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  PLK2 c.328G>A |  |  |  | -50.0 [-90.5 to 48.6]
  PLXNA1 c.1114C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  PLXNA1 c.1114C>T |  |  |  | -50.0 [-90.5 to 48.6]
  PLXND1 c.1393G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  PLXND1 c.1393G>A |  |  |  | 50.0 [-48.6 to 90.5]
  PML c.1753delC: number analyzed (Participants) | 0 | 0 | 0 | 2
  PML c.1753delC |  |  |  | -50.0 [-90.5 to 48.6]
  PODXL2 c.1230delG: number analyzed (Participants) | 0 | 0 | 0 | 2
  PODXL2 c.1230delG |  |  |  | -50.0 [-90.5 to 48.6]
  POLQ c.6811C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  POLQ c.6811C>A |  |  |  | -50.0 [-90.5 to 48.6]
  POLR2B c.632delA: number analyzed (Participants) | 0 | 0 | 0 | 2
  POLR2B c.632delA |  |  |  | -50.0 [-90.5 to 48.6]
  POM121 c.1916A>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  POM121 c.1916A>C |  |  |  | 50.0 [-48.6 to 90.5]
  POM121C c.1162_1169delTTTGACTCinsCT: number analyzed (Participants) | 0 | 0 | 0 | 2
  POM121C c.1162_1169delTTTGACTCinsCT |  |  |  | 0.0 [-65.8 to 65.8]
  POTEB2 c.119C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  POTEB2 c.119C>A |  |  |  | 50.0 [-48.6 to 90.5]
  PPP1R12C c.1907C>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  PPP1R12C c.1907C>G |  |  |  | -50.0 [-90.5 to 48.6]
  PPP2R2B c.1196G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  PPP2R2B c.1196G>A |  |  |  | 50.0 [-48.6 to 90.5]
  PPWD1 c.197-6_198delCTTCAGTCinsTTTTTTTT: number analyzed (Participants) | 0 | 0 | 0 | 2
  PPWD1 c.197-6_198delCTTCAGTCinsTTTTTTTT |  |  |  | 50.0 [-48.6 to 90.5]
  PRAMEF2 c.280C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  PRAMEF2 c.280C>T |  |  |  | -50.0 [-90.5 to 48.6]
  PRKDC c.2601C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  PRKDC c.2601C>A |  |  |  | 50.0 [-48.6 to 90.5]
  PROSER1 c.1587G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  PROSER1 c.1587G>T |  |  |  | -50.0 [-90.5 to 48.6]
  PRR19 c.355C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  PRR19 c.355C>T |  |  |  | 50.0 [-48.6 to 90.5]
  PRRT3 c.543G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  PRRT3 c.543G>T |  |  |  | -50.0 [-90.5 to 48.6]
  PRSS56 c.1646G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  PRSS56 c.1646G>A |  |  |  | -50.0 [-90.5 to 48.6]
  PTPN13 c.4093G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  PTPN13 c.4093G>T |  |  |  | -50.0 [-90.5 to 48.6]
  R3HDM2 c.79_80delAA: number analyzed (Participants) | 0 | 0 | 0 | 2
  R3HDM2 c.79_80delAA |  |  |  | 0.0 [-65.8 to 65.8]
  RABGEF1 c.854C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  RABGEF1 c.854C>T |  |  |  | -50.0 [-90.5 to 48.6]
  RAD50 c.2165delA: number analyzed (Participants) | 0 | 0 | 0 | 2
  RAD50 c.2165delA |  |  |  | -50.0 [-90.5 to 48.6]
  RAP2B c.56T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  RAP2B c.56T>G |  |  |  | 0.0 [-65.8 to 65.8]
  RASGEF1A c.1062delC: number analyzed (Participants) | 0 | 0 | 0 | 2
  RASGEF1A c.1062delC |  |  |  | 0.0 [-65.8 to 65.8]
  RBM15 c.1231G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  RBM15 c.1231G>A |  |  |  | -50.0 [-90.5 to 48.6]
  RBMX c.217-2_217-1delAGinsTT: number analyzed (Participants) | 0 | 0 | 0 | 2
  RBMX c.217-2_217-1delAGinsTT |  |  |  | 50.0 [-48.6 to 90.5]
  RD3 c.292C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  RD3 c.292C>T |  |  |  | -50.0 [-90.5 to 48.6]
  RGPD1 c.4329A>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  RGPD1 c.4329A>C |  |  |  | 50.0 [-48.6 to 90.5]
  RGS17 c.55C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  RGS17 c.55C>T |  |  |  | 0.0 [-65.8 to 65.8]
  RIMBP2 c.2627C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  RIMBP2 c.2627C>T |  |  |  | 0.0 [-65.8 to 65.8]
  RLBP1 c.307C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  RLBP1 c.307C>T |  |  |  | 0.0 [-65.8 to 65.8]
  RNF128 c.103G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  RNF128 c.103G>A |  |  |  | -50.0 [-90.5 to 48.6]
  RRN3 c.337A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  RRN3 c.337A>G |  |  |  | 50.0 [-48.6 to 90.5]
  RSL1D1 c.1147-5_1147delCTTAGAinsTTTTTT: number analyzed (Participants) | 0 | 0 | 0 | 2
  RSL1D1 c.1147-5_1147delCTTAGAinsTTTTTT |  |  |  | 50.0 [-48.6 to 90.5]
  RSPH3 c.1186G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  RSPH3 c.1186G>A |  |  |  | 0.0 [-65.8 to 65.8]
  RTTN c.5365G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  RTTN c.5365G>A |  |  |  | -50.0 [-90.5 to 48.6]
  S100A7 c.139T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  S100A7 c.139T>G |  |  |  | 0.0 [-65.8 to 65.8]
  SAMD13 c.169G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SAMD13 c.169G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SCML2 c.654G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  SCML2 c.654G>T |  |  |  | -50.0 [-90.5 to 48.6]
  SCN1A c.1363C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SCN1A c.1363C>A |  |  |  | 0.0 [-65.8 to 65.8]
  SCN7A c.2098G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SCN7A c.2098G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SCRIB c.4063C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  SCRIB c.4063C>T |  |  |  | 50.0 [-48.6 to 90.5]
  SDK1 c.1769C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SDK1 c.1769C>A |  |  |  | -50.0 [-90.5 to 48.6]
  SDK2 c.4706C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SDK2 c.4706C>A |  |  |  | -50.0 [-90.5 to 48.6]
  SEC24A c.2346C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SEC24A c.2346C>A |  |  |  | -50.0 [-90.5 to 48.6]
  SEMA6D c.509C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  SEMA6D c.509C>T |  |  |  | -50.0 [-90.5 to 48.6]
  SESN1 c.1469G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SESN1 c.1469G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SFT2D3 c.314C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  SFT2D3 c.314C>T |  |  |  | -50.0 [-90.5 to 48.6]
  SHANK1 c.1329G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  SHANK1 c.1329G>T |  |  |  | -50.0 [-90.5 to 48.6]
  SHANK1 c.1366G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SHANK1 c.1366G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SHROOM2 c.2815C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SHROOM2 c.2815C>A |  |  |  | -50.0 [-90.5 to 48.6]
  SIX3 c.406_407delGC: number analyzed (Participants) | 0 | 0 | 0 | 2
  SIX3 c.406_407delGC |  |  |  | -50.0 [-90.5 to 48.6]
  SLC30A10 c.1408C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SLC30A10 c.1408C>A |  |  |  | -50.0 [-90.5 to 48.6]
  SPTBN5 c.2405G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SPTBN5 c.2405G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SPTLC1 c.1110C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SPTLC1 c.1110C>A |  |  |  | -50.0 [-90.5 to 48.6]
  ST7 c.1658G>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  ST7 c.1658G>C |  |  |  | -50.0 [-90.5 to 48.6]
  STARD9 c.1654C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  STARD9 c.1654C>T |  |  |  | 50.0 [-48.6 to 90.5]
  STK32A c.326G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  STK32A c.326G>A |  |  |  | 0.0 [-65.8 to 65.8]
  STRBP c.709C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  STRBP c.709C>T |  |  |  | 0.0 [-65.8 to 65.8]
  SVIL c.2083G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SVIL c.2083G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SYNE1 c.23551A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  SYNE1 c.23551A>G |  |  |  | 50.0 [-48.6 to 90.5]
  SYNGR1 c.34G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SYNGR1 c.34G>A |  |  |  | 50.0 [-48.6 to 90.5]
  TACC2 c.798G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  TACC2 c.798G>T |  |  |  | -50.0 [-90.5 to 48.6]
  TCF7L1 c.40_42delGGC: number analyzed (Participants) | 0 | 0 | 0 | 2
  TCF7L1 c.40_42delGGC |  |  |  | 50.0 [-48.6 to 90.5]
  TCTN2 c.127G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  TCTN2 c.127G>A |  |  |  | 0.0 [-65.8 to 65.8]
  TEX30 c.132_133delTC: number analyzed (Participants) | 0 | 0 | 0 | 2
  TEX30 c.132_133delTC |  |  |  | -50.0 [-90.5 to 48.6]
  TFCP2L1 c.161C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  TFCP2L1 c.161C>T |  |  |  | -50.0 [-90.5 to 48.6]
  TM4SF1 c.199T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  TM4SF1 c.199T>G |  |  |  | 0.0 [-65.8 to 65.8]
  TMEM202 c.603C>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  TMEM202 c.603C>G |  |  |  | 0.0 [-65.8 to 65.8]
  TMEM26 c.709G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  TMEM26 c.709G>T |  |  |  | -50.0 [-90.5 to 48.6]
  TMEM72 c.490G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  TMEM72 c.490G>A |  |  |  | -50.0 [-90.5 to 48.6]
  TMOD3 c.151C>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  TMOD3 c.151C>G |  |  |  | 0.0 [-65.8 to 65.8]
  TMPO c.514A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  TMPO c.514A>G |  |  |  | 0.0 [-65.8 to 65.8]
  TMPRSS6 c.435C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  TMPRSS6 c.435C>A |  |  |  | -50.0 [-90.5 to 48.6]
  SKP1 c.21G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  SKP1 c.21G>T |  |  |  | -50.0 [-90.5 to 48.6]
  SLC25A12 c.887C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SLC25A12 c.887C>A |  |  |  | -50.0 [-90.5 to 48.6]
  SLC2A11 c.995C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  SLC2A11 c.995C>T |  |  |  | -50.0 [-90.5 to 48.6]
  SLC35F2 c.448G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SLC35F2 c.448G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SLC38A2 c.549T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  SLC38A2 c.549T>G |  |  |  | 0.0 [-65.8 to 65.8]
  SLC39A6 c.1088C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  SLC39A6 c.1088C>T |  |  |  | -50.0 [-90.5 to 48.6]
  SLC5A2 c.236G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SLC5A2 c.236G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SLC7A14 c.1963T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  SLC7A14 c.1963T>C |  |  |  | 0.0 [-65.8 to 65.8]
  SLC7A9 c.887G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SLC7A9 c.887G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SLU7 c.576delA: number analyzed (Participants) | 0 | 0 | 0 | 2
  SLU7 c.576delA |  |  |  | 50.0 [-48.6 to 90.5]
  SOAT1 c.1421T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  SOAT1 c.1421T>G |  |  |  | 50.0 [-48.6 to 90.5]
  SOCS6 c.781G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SOCS6 c.781G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SORBS1 c.3400G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SORBS1 c.3400G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SP140 c.205G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  SP140 c.205G>T |  |  |  | -50.0 [-90.5 to 48.6]
  SPATA31E1 c.2651G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  SPATA31E1 c.2651G>A |  |  |  | -50.0 [-90.5 to 48.6]
  SPPL2B c.634G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  SPPL2B c.634G>T |  |  |  | -50.0 [-90.5 to 48.6]
  TMPRSS6 c.943G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  TMPRSS6 c.943G>A |  |  |  | -50.0 [-90.5 to 48.6]
  TNFAIP2 c.512_514delCGG: number analyzed (Participants) | 0 | 0 | 0 | 2
  TNFAIP2 c.512_514delCGG |  |  |  | 50.0 [-48.6 to 90.5]
  TNXB c.8806G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  TNXB c.8806G>A |  |  |  | -50.0 [-90.5 to 48.6]
  TOGARAM2 c.2090C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  TOGARAM2 c.2090C>A |  |  |  | -50.0 [-90.5 to 48.6]
  TOP3B c.2299T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  TOP3B c.2299T>C |  |  |  | 50.0 [-48.6 to 90.5]
  TRIM17 c.232C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  TRIM17 c.232C>T |  |  |  | 0.0 [-65.8 to 65.8]
  TRIM28 c.335G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  TRIM28 c.335G>A |  |  |  | -50.0 [-90.5 to 48.6]
  TRIM3 c.2235G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  TRIM3 c.2235G>T |  |  |  | 0.0 [-65.8 to 65.8]
  TRIO c.9289G>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  TRIO c.9289G>C |  |  |  | 0.0 [-65.8 to 65.8]
  TRIP12 c.1099C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  TRIP12 c.1099C>T |  |  |  | -50.0 [-90.5 to 48.6]
  TSHZ1 c.1204G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  TSHZ1 c.1204G>A |  |  |  | -50.0 [-90.5 to 48.6]
  TSPEAR c.59C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  TSPEAR c.59C>T |  |  |  | -50.0 [-90.5 to 48.6]
  TSSC4 c.538G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  TSSC4 c.538G>T |  |  |  | 0.0 [-65.8 to 65.8]
  TVP23A c.271T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  TVP23A c.271T>C |  |  |  | 50.0 [-48.6 to 90.5]
  UBD c.3G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  UBD c.3G>A |  |  |  | -50.0 [-90.5 to 48.6]
  UBE2O c.1813G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  UBE2O c.1813G>A |  |  |  | -50.0 [-90.5 to 48.6]
  UGDH c.1294delA: number analyzed (Participants) | 0 | 0 | 0 | 2
  UGDH c.1294delA |  |  |  | -50.0 [-90.5 to 48.6]
  UGGT2 c.3474-467_3480del: number analyzed (Participants) | 0 | 0 | 0 | 2
  UGGT2 c.3474-467_3480del |  |  |  | 50.0 [-48.6 to 90.5]
  URI1 c.49G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  URI1 c.49G>T |  |  |  | -50.0 [-90.5 to 48.6]
  USP28 c.2845C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  USP28 c.2845C>T |  |  |  | 50.0 [-48.6 to 90.5]
  USP34 c.1142C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  USP34 c.1142C>A |  |  |  | -50.0 [-90.5 to 48.6]
  UTF1 c.302C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  UTF1 c.302C>T |  |  |  | -50.0 [-90.5 to 48.6]
  VSTM2B c.457G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  VSTM2B c.457G>A |  |  |  | 50.0 [-48.6 to 90.5]
  VSTM2B c.603C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  VSTM2B c.603C>A |  |  |  | -50.0 [-90.5 to 48.6]
  WASHC2C c.1562A>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  WASHC2C c.1562A>C |  |  |  | 50.0 [-48.6 to 90.5]
  WASHC2C c.691G>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  WASHC2C c.691G>T |  |  |  | -50.0 [-90.5 to 48.6]
  WDR33 c.160C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  WDR33 c.160C>T |  |  |  | -50.0 [-90.5 to 48.6]
  WFS1 c.577_579delAAG: number analyzed (Participants) | 0 | 0 | 0 | 2
  WFS1 c.577_579delAAG |  |  |  | -50.0 [-90.5 to 48.6]
  WISP1 c.580A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  WISP1 c.580A>G |  |  |  | -50.0 [-90.5 to 48.6]
  WWC1 c.2972T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  WWC1 c.2972T>G |  |  |  | 0.0 [-65.8 to 65.8]
  YBX3 c.40_42delACC: number analyzed (Participants) | 0 | 0 | 0 | 2
  YBX3 c.40_42delACC |  |  |  | 50.0 [-48.6 to 90.5]
  ZFPM1 c.2596C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZFPM1 c.2596C>T |  |  |  | -50.0 [-90.5 to 48.6]
  ZNF148 c.2380_2383delGGCTinsAA: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF148 c.2380_2383delGGCTinsAA |  |  |  | 50.0 [-48.6 to 90.5]
  ZNF185 c.1222G>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF185 c.1222G>A |  |  |  | -50.0 [-90.5 to 48.6]
  ZNF221 c.335C>T: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF221 c.335C>T |  |  |  | 50.0 [-48.6 to 90.5]
  ZNF354C c.1060A>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF354C c.1060A>G |  |  |  | 50.0 [-48.6 to 90.5]
  ZNF366 c.1475T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF366 c.1475T>G |  |  |  | 0.0 [-65.8 to 65.8]
  ZNF41 c.1700_1702delAAA: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF41 c.1700_1702delAAA |  |  |  | 0.0 [-65.8 to 65.8]
  ZNF521 c.3122T>C: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF521 c.3122T>C |  |  |  | 0.0 [-65.8 to 65.8]
  ZNF550 c.157C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF550 c.157C>A |  |  |  | -50.0 [-90.5 to 48.6]
  ZNF552 c.524_525dupGG: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF552 c.524_525dupGG |  |  |  | 50.0 [-48.6 to 90.5]
  ZNF552 c.533T>G: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF552 c.533T>G |  |  |  | 50.0 [-48.6 to 90.5]
  ZNF628 c.794C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF628 c.794C>A |  |  |  | -50.0 [-90.5 to 48.6]
  ZNF883 c.664C>A: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZNF883 c.664C>A |  |  |  | 0.0 [-65.8 to 65.8]
  ZSWIM6 c.82_84dupAGC: number analyzed (Participants) | 0 | 0 | 0 | 2
  ZSWIM6 c.82_84dupAGC |  |  |  | 50.0 [-48.6 to 90.5]

2. Secondary Outcome: Number of Participants With Fully Evaluable Archival and Post-Progression Tumor Biopsy by Cohort
Description: Estimating the number of fully biomarker evaluable population by cohort to evaluate the success rate in obtaining paired archival and post-progression tumor biopsies that were adequate to meet the objectives of the study
Time Frame: Through study completion, approximately 3 months
Population: Participants included in the Safety Analysis population in 7 cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: NSCLC Monotherapy | Cohort 2: NSCLC Combination | Cohort 3: RCC With Clear Cell Component | Cohort 4: HR+ HER2- Adenocarcinoma of the Breast | Cohort 5: Castrate-resistant Adenocarcinoma of the Prostate | Cohort 6: Castrate-resistant Adenocarcinoma of the Prostate | Cohort 7: gBRCAm HER2- Adenocarcinoma of the Breast
Number analyzed (Participants) | 1 | 4 | 5 | 11 | 5 | 11 | 1
Participants
  Safety Analysis (SA) | 1 | 4 | 5 | 10 | 5 | 10 | 1
  Biomarker Evaluable (BE) | 1 | 4 | 5 | 8 | 5 | 8 | 1
  Biomarker Evaluable Target (BET) | 0 | 1 | 3 | 6 | 4 | 2 | 1
  Fully Biomarker Evaluable (FBE) | 0 | 1 | 1 | 1 | 1 | 0 | 0

3. Secondary Outcome: Overall Agreement Rate of Gene Alterations Between Post-Progression Tumor Biopsy and Blood NGS Results
Description: Genetic alterations detected in blood were compared to those detected in tissue. Only gene alterations with frequency of 5% or greater based on assessment of tumor biopsy were included in the analysis.
Time Frame: Through study completion, approximately 3 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Percentage of agreed gene alterations
Groups:
- HR+HER2-adenocarcinoma of the Breast (Cohort 4): Progressive disease on 1st line combination of doublet palbociclib with hormonal therapy.
- Castrate-resistant Adenocarcinoma of the Prostate (Cohort 5 & 6): Progressive disease on enzalutamide monotherapy and on abiraterone in combination with prednisone.
Arm/Group | HR+HER2-adenocarcinoma of the Breast (Cohort 4) | Castrate-resistant Adenocarcinoma of the Prostate (Cohort 5 & 6)
Number analyzed (Participants) | 8 | 10
Percentage of agreed gene alterations | 11.9 [0.0 to 18.8] | 0.0 [0.0 to 16.7]

4. Secondary Outcome: Change in Frequency of RB1 Gene Alterations Between Pre-Treatment Archival and Post-Progression Samples
Description: Mutations in RB1 gene associated with immune function, have also been shown to impact tumor immunogenicity and related with CDK4/6 inhibition. CDK4 or CDK6 complexed with cyclin D1 (CCND1) phosphorylates the retinoblastoma gene product (Rb), releasing the E2F and DP transcription factors that regulate the expression of genes required for entry into the S phase of the cell cycle.
  Calculation of change in frequency was decribed in the primary endpoint (Outcome Measure 1).
Time Frame: Through study completion, approximately 3 months
Population: The BET population was participants in the BE population who had a targeted tumor DNA panel biomarker result from both archival and de novo biopsy tumor tissue biospecimen. BET (WETD) was defined as all participants in the BET population who had results of WETD NGS sample analysis from both the archival and de novo biopsy tumor tissue biospecimen. RB1 Gene Alterations analysis was only conducted for Cohort 4 as per protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- HR+HER2-adenocarcinoma of the Breast in the BET Populations (Cohort 4); HR+HER2-adenocarcinoma of the Breast in the BET (WETD) Populations (Cohort 4): Progressive disease on 1st line combination of doublet palbociclib with hormonal therapy.
Arm/Group | HR+HER2-adenocarcinoma of the Breast in the BET Populations (Cohort 4) | HR+HER2-adenocarcinoma of the Breast in the BET (WETD) Populations (Cohort 4)
Number analyzed (Participants) | 6 | 3
Percentage of participants | 0.0 [-39.0 to 39.0] | -33.3 [-79.2 to 41.5]

5. Secondary Outcome: Percentage of Participants Who Carried the RB1 Gene Alterations in Post-Progression Blood cfDNA
Description: Mutations in RB1 gene associated with immune function, have also been shown to impact tumor immunogenicity and related with CDK4/6 inhibition. CDK4 or CDK6 complexed with cyclin D1 (CCND1) phosphorylates the retinoblastoma gene product (Rb), releasing the E2F and DP transcription factors that regulate the expression of genes required for entry into the S phase of the cell cycle. Percentage of Participants Who Carried the RB1 Gene Alterations in Post Progression Blood cfDNA analysis was only conducted for Cohort 4 as per protocol.
Time Frame: Through study completion, approximately 3 months
Population: BE (TBD) was analyzed and defined as all participants in the BE population who have results of targeted blood cfDNA (TBD) NGS gene panel sample analysis from the post-progression blood sample.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- HR+HER2-adenocarcinoma of the Breast in the BE (TBD) Populations (Cohort 4): Progressive disease on 1st line combination of doublet palbociclib with hormonal therapy.
Arm/Group | HR+HER2-adenocarcinoma of the Breast in the BE (TBD) Populations (Cohort 4)
Number analyzed (Participants) | 8
Percentage of participants
  c.151G>T | 12.5 [2.2 to 47.1]
  c.184C>T | 12.5 [2.2 to 47.1]
  c.54_79delGGAACCCCCGGCACCGCCGCCGCCGC | 12.5 [2.2 to 47.1]

6. Secondary Outcome: Change in Frequency of AR Gene Alterations Between Pre-Treatment Archival and Post-Progression Samples
Description: Pre-treatment archival tumor samples and post-progression de novo tumor biopsies were analyzed to identify molecular markers of resistance to selected anti-cancer therapies.
  Calculation of change in frequency was described for in the primary endpoint (Outcome Measure 1).
  AR gene Alterations analysis was only conducted for the Cohorts 5 & 6 as per protocol.
Time Frame: Through study completion, approximately 3 months
Population: The BET and BET (WETD) population was participants in the BE population who have a targeted tumor DNA panel biomarker result, and all participants in the BET population who have results of WETD NGS sample analysis, from both the archival and de novo biopsy tumor tissue biospecimen, respectively. One participant in Cohort 6 was included in the BET analysis population given the small number of eligible samples and the fact that participant's bone sample met analytical requirements.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Castrate-resistant Adenocarcinoma of the Prostate in the BET Populations (Cohort 5 & 6); Castrate-resistant Adenocarcinoma of the Prostate in the BET (WETD) Populations (Cohort 5 & 6): Progressive disease on enzalutamide monotherapy and on abiraterone in combination with prednisone.
Arm/Group | Castrate-resistant Adenocarcinoma of the Prostate in the BET Populations (Cohort 5 & 6) | Castrate-resistant Adenocarcinoma of the Prostate in the BET (WETD) Populations (Cohort 5 & 6)
Number analyzed (Participants) | 6 | 2
percentage of participants | 0.0 [-39.0 to 39.0] | 0.0 [-65.8 to 65.8]

7. Secondary Outcome: Percentage of Participants Who Carried the AR Gene Alterations in Post-Progression Blood cfDNA
Description: Androgen receptor (AR) gene alterations can be evaluated as mechanisms of resistance to enzalutamide or abiraterone.
  Percentage of Participants Who Carried the AR Gene Alterations in Post-Progression Blood cfDNA analysis was conducted as it was only applicable to Cohorts 5 &6.
Time Frame: Through study completion, approximately 3 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Castrate-resistant Adenocarcinoma of the Prostate in the BE (TBD) Populations (Cohort 5 & 6): Progressive disease on enzalutamide monotherapy and on abiraterone in combination with prednisone.
Arm/Group | Castrate-resistant Adenocarcinoma of the Prostate in the BE (TBD) Populations (Cohort 5 & 6)
Number analyzed (Participants) | 10
Percentage of participants
  c.2105T>A | 20.0 [5.7 to 51.0]
  c.2202G>C | 10.0 [1.8 to 40.4]
  c.2632A>G | 10.0 [1.8 to 40.4]

8. Secondary Outcome: Change in Expression of Nuclear Hormone Receptors Between Pre-Treatment Archival and Post-Progression Samples
Description: The differences in the expression of nuclear hormone receptor (HR) reflecting nuclear receptor pathway activity between the archival and de novo samples. Using HTG panel in BET [targeted tumor RNA (TTR)] population and Tempus RNAseq in BET [whole transcriptome tumor RNA (WTTR)] population. The unit of HTG expression data for nuclear hormone receptors is normalized expression counts. This Outcome Measure analysis was only conducted for Cohorts 5 & 6 as per protocol.
Time Frame: Through study completion, approximately 3 months
Population: BET (TTR) and BET (WTTR) population was all participants in the BET population who have results of TTR sample analysis, and all participants in the BET population who have results of WTTR NGS sample analysis, from both the archival and de novo biopsy tumor tissue biospecimen, respectively. One participant in Cohort 6 was included in the BET analysis population given the small number of eligible samples and the fact that participant's bone sample met analytical requirements.
Measure: Mean (95% Confidence Interval); unit: normalized expression counts
Groups:
- Castrate-resistant Adenocarcinoma of the Prostate in the BET (TTR) Populations (Cohort 5 & 6); Castrate-resistant Adenocarcinoma of the Prostate in the BET (WTTR) Populations (Cohort 5 & 6): Progressive disease on enzalutamide monotherapy and on abiraterone in combination with prednisone.
Arm/Group | Castrate-resistant Adenocarcinoma of the Prostate in the BET (TTR) Populations (Cohort 5 & 6) | Castrate-resistant Adenocarcinoma of the Prostate in the BET (WTTR) Populations (Cohort 5 & 6)
Number analyzed (Participants) | 2 | 6
normalized expression counts
  ESR1 | 0.3 [-16.4 to 17.1] | 25.6 [-11.2 to 62.5]
  ESR2 | -0.4 [-6.3 to 5.5] | -1.1 [-2.3 to 0.1]
  NR3C1 | 0.5 [-1.2 to 2.1] | 5.4 [-30.7 to 41.5]
  NR3C2: number analyzed (Participants) | 0 | 6
  NR3C2 |  | 3.7 [-18.2 to 25.6]
  PGR | -0.5 [-13.4 to 12.4] | 2.0 [-3.9 to 7.9]
  AR | -0.7 [-10.9 to 9.4] | 549.9 [-480.1 to 1579.9]

ADVERSE EVENTS:
Time Frame: From Biospecimen Collection Day 1 to Post-Biospecimen Follow-up ≤30 days after receipt of NGS results at the provider's facility, approximately 3 months through study completion.
Arm/Group | Cohort 1: NSCLC Monotherapy | Cohort 2: NSCLC Combination | Cohort 3: RCC With Clear Cell Component | Cohort 4: HR+ HER2- Adenocarcinoma of the Breast | Cohort 5: Castrate-resistant Adenocarcinoma of the Prostate | Cohort 6: Castrate-resistant Adenocarcinoma of the Prostate | Cohort 7: gBRCAm HER2- Adenocarcinoma of the Breast
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4 | 0/5 | 0/10 | 0/5 | 0/10 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4 | 0/5 | 0/10 | 0/5 | 0/10 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4 | 0/5 | 1/10 | 1/5 | 0/10 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: NSCLC Monotherapy (N=1) | Cohort 2: NSCLC Combination (N=4) | Cohort 3: RCC With Clear Cell Component (N=5) | Cohort 4: HR+ HER2- Adenocarcinoma of the Breast (N=10) | Cohort 5: Castrate-resistant Adenocarcinoma of the Prostate (N=5) | Cohort 6: Castrate-resistant Adenocarcinoma of the Prostate (N=10) | Cohort 7: gBRCAm HER2- Adenocarcinoma of the Breast (N=1)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Because of given challenges with study enrollment that were compounded by the global COVID-19 pandemic, and the observed high failure rate of tumor biospecimen analyses due to limitations in sample quality and quantity, the study was terminated in October 2020, which was not due to safety concerns or regulatory interactions. For endpoints with no data collected, no results can be disclosed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT04436120/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT04436120/SAP_001.pdf